#### **PrEP Protocol Outline**

## August 30, 2023

AURORA Study-A Transformative Approach Utilizing Behavioral Economics, Education, and Data Science to Support Patients Initiating PrEP with Retention-in-care and Medication Persistence

Cover Page with signature page

**Protocol Team** 

W. David Hardy, MD, AAHIVS (Principal Investigator)
Adjunct Clinical Professor of Medicine
Division of Infectious Diseases
Keck School of Medicine of USC

Angie Settle, DNP, APRN,BC, FNP CEO, WV Health Right

Kelly Pillinger, PharmD, BCPS, BCIDP

PRIME Education, LLC

Kelly & Pillinger

Jeffrey Carter, PhD PRIME Education, LLC

Jall Carrie

## **List of Abbreviations**

- CAB-LA Long-Acting Injectable Cabotegravir
- EHR Electronic Health Record
- FTC Emtricitabine
- TDF Tenofovir disoproxil
- TAF Tenofovir alafenamide
- HCP Health Care Provider
- HIV Human Immunodeficiency Virus
- PrEP Pre-Exposure Prophylaxis
- PROs Patient Reported Outcomes
- PWID Persons who inject drugs
- WVHR West Virginia Health Right

## 1. PROTOCOL SUMMARY

| Title | A Transformative Approach Utilizing Behavioral Economics, Education, |
|---|---|
| | and Data Science to Support Patients Initiating PrEP with Retention-in- |
| | care and Medication Adherence and Persistence |
| Funder | ViiV Healthcare |
| Study Design | Observational Cohort Study |
| Study Population | Patients >18 y/o who are newly started on PrEP at WVHR and have |
| | access to a smart phone with data. |
| Study Size | n = 105 (70 CAB-LA injection participants and |
| | 35 oral PrEP participants) |

| Study Duration | 12 months |
|---|---|
| Study Site(s) | West Virginia Health Right |
| Intervention | Participants will have been prescribed CAB-LA, daily FTC/TDF, or daily |
| Description | FTC/TAF in accordance with the WVHR standard of care by a licensed |
| | HCP prior to enrolling in the study. Those receiving CAB-LA will be in |
| | one arm and those receiving oral PrEP will be in the other arm of the |
| | study. |
| Study Aim | To determine the persistence of injectable PrEP compared to oral PrEP |
| Primary Objectives | To evaluate medication persistence in patients receiving CAB-LA |
| | injections vs oral PrEP and who engage with a digital health |
| | companion program |
| Secondary | Evaluate retention-in-care in patients receiving CAB-LA vs oral |
| Objective 1 | PrEP |
| Secondary | Evaluate PROs (including PrEP medication satisfaction, PrEP |
| Objective 2 | acceptance, PrEP-Related Stigma, and reasons for PrEP |
| | discontinuation) in patients receiving CAB-LA vs oral PrEP |
| Secondary | Evaluate the acceptability, appropriateness, and helpfulness of a |
| Objective 3 | digital health companion program for PrEP |
| Secondary | Evaluate the acceptability, barriers to, and facilitators for |
| Objective 4 | implementation of CAB-LA PrEP |

## 2. INTRODUCTION

## 2.1. Background

2.1.1. Numerous studies have found that medication persistence with oral PrEP (defined as continued use of PrEP over time) tends to be short, with many patients discontinuing oral PrEP within about 6-12 months. Moreover, PrEP persistence has been found to be shorter among underserved populations with heath inequities—including Medicaid patients, patients in rural areas, transgender patients, and Black and Latinx patients. The introduction of long-acting, injectable cabotegravir (CABLA) for PrEP is viewed by many as an opportunity to overcome adherence

challenges. Moreover, based on its administration by a healthcare professional (HCP) every two months, the implementation for CAB-LA in real-world settings affords HCPs new opportunities to engage with patients, especially those with high unmet needs, which may influence PrEP persistence, retention-in-care, and patient-reported outcomes (PROs). To support adoption of CAB-LA for HIV PrEP, real-world studies are urgently needed to evaluate the impact of CAB-LA on outcomes that are critical to successful HIV prevention, such as adherence, persistence, retention-in-care, and PROs. Additionally, given its mode of administration, studies are needed to elucidate barriers to as well as facilitators for the implementation of CAB-LA PrEP in clinical settings. For people living with HIV, findings from the CUSTOMIZE study shed light on patient and provider perspectives on implementation of CAB+RPV LA for treatment of HIV. These insights from diverse settings of HIV treatment can serve as a springboard for evidence generation on the real-world use of CAB-LA for PrEP. Recognizing the need to support clinics in implementing and streamlining the delivery of PrEP, PRIME recently partnered with West Virginia Health Right (WVHR) in an implementation science initiative. Through this initiative, significant advances were made in overcoming barriers related to PrEP access. Specifically, the initiative directly resulted in a landmark decision by the Director of the West Virginia Medicaid program to remove all prior authorization requirements for CAB-LA for PrEP after attending the PRIME program. Building on this momentum and reduced barriers to CAB-LA access in WV, we propose to evaluate the implementation of CAB-LA supported by a novel PrEP mobile health app among underserved populations receiving care at WVHR. WVHR is a 501(c)3 non-profit, patientcentered, medical home that provides comprehensive primary and specialty care to >40,000 uninsured, underinsured, and underserved adults. Among services provided, WVHR provides HIV prevention care, harm reduction services, behavioral health care, and transgender health care—which is the only transgender health program in the region. Its in-house pharmacy fills >90,000 prescriptions annually,

including access to free medications for uninsured patients. Additionally, WVHR utilizes a mobile health clinic to care for hard-to-reach populations. WVHR is in Kanawha County, which is designated by the CDC as one of the top vulnerable areas of rapid spread of HIV due to injection drug use. Due to its location, services provided, and focus on uninsured/underinsured individuals, the populations cared for by WVHR encompass those with high unmet needs and PrEP-related disparities, including women, persons who inject drugs (PWID), transgender persons, persons in rural areas, and persons with low-income. Importantly, WVHR is committed to sustaining the HIV prevention initiative after the proposed study has concluded, as stated in the letter from Chief Executive Officer, Angie Settle, DNP, APRN, BC, FNP

## 2.2. Study Rationale

2.2.1. The digital health companion intervention that will be utilized in this research project is based on combining the principles of behavioral health economics, patient education, and data science to drive positive behavior change in PrEP adherence, persistence and retention-in-care. Prior research supports the acceptability and effectiveness of mobile health interventions for adherence to oral PrEP. For example, a PrEP adherence mobile app ("Dot"), which was tailored for culturally-diverse MSM, was found to have high user acceptability and resulted in increased adherence to daily PrEP over the 6-week intervention. Other mobile interventions have similarly been found to be effective in supporting PrEP adherence in key populations, including in MSM (PrEPmate, Viral combat) and cisgender women (AEGiS/iTAB). Importantly, surveys show that 86% of Medicaid beneficiaries own smartphones and that approximately one-quarter to one-half use their smartphone for a variety of health purposes, such as filling prescriptions, measuring health goals, monitoring health issues, and receiving reminders about prescription drugs. Thus, there is an important opportunity to evaluate mobile health interventions for PrEP among low-income, Medicaid populations, and to expand the use of mobile interventions for supporting persistence to long-acting injectable PrEP.

## 2.3. Hypothesis

2.3.1. This study is designed to test the hypothesis that, compared to oral PrEP, use of CAB-LA in underserved populations in a real-world setting supported by a digital health companion program will be associated with greater medication adherence, persistence, retention-in-care, and improved PROs.

## 3. STUDY OBJECTIVES

## 3.1. Study Goal

3.1.1. The study will evaluate the extent to which real-world use of CAB-LA for PrEP in underserved populations impacts PrEP adherence, persistence, retention-in-care, and PROs compared with oral PrEP. Additionally, the study will examine implementation of a digital health companion program that leverages education and behavioral economics to support patients on PrEP, and assess clinician perspectives as well as barriers to, and facilitators for implementation of CAB-LA in a patient-centered medical home.

## 3.2. Primary Objective

3.2.1. To evaluate medication adherence and persistence in patients receiving CAB-LA vs oral PrEP and who engage with a digital health companion program

## 3.3. Secondary Objectives

- 3.3.1. Evaluate retention-in-care in patients receiving CAB-LA vs oral PrEP
- 3.3.2. Evaluate PROs (including PrEP Medication Satisfaction, PrEP Acceptance, PrEP-Related Stigma, and reasons for PrEP discontinuation) in patients receiving CAB-LA vs oral PrEP
- 3.3.3. Evaluate the acceptability, appropriateness, and helpfulness of a digital health companion program for PrEP
- 3.3.4. Evaluate the acceptability, barriers to, and facilitators for implementation of CAB-LA

#### 4. STUDY DESIGN

4.1. Study Design

4.1.1. The research project follows a hybrid effectiveness-implementation research design, with the primary aim focused on evaluation of PrEP adherence, persistence and retention-in-care with CAB-LA compared with oral PrEP, and secondary aims focused on evaluating patient-reported outcomes (PROs), implementation of a digital health intervention to support adherence and persistence, and evaluating contextual factors around implementation of CAB-LA. The project is in the initial implementation stage, with CAB-LA beginning to be rolled out at WVHR after the recent state Medicaid decision to drop prior authorization requirements for CAB-LA. The proposed study will utilize a digital health intervention with behavioral health economics and patient education from PRIME and Reciprocity to evaluate the adoption and implementation for PrEP adherence and persistence. The implementation aims of the study will leverage the RE-AIM framework as follows: Assessment of the digital health intervention will focus primarily on individual-level dimensions of RE-AIM, including reach and effectiveness. For example, in assessing reach of the digital health intervention, participant demographics will be compared to the intended audience to evaluate the extent to which populations with high unmet needs were engaged. Conversely, assessment of the implementation of CAB-LA will focus on system-level dimensions of RE-AIM, such as qualitative assessments of barriers to and facilitators for implementation of CAB-LA. Furthermore, evaluation of implementation outcomes will be based on the Proctor et al. conceptual framework, using specific measures developed by Weiner et al. to assess acceptability, appropriateness, and feasibility of the intervention. In addition, evaluation of PROs will be informed by a review of validated instruments, including HIVSTQ (HIV Treatment Satisfaction Questionnaire), SMSQ (Study Medication Satisfaction Questionnaire), I-TAQ (Injection Treatment Acceptance Questionnaire), ACCEPT (Chronic Treatment Acceptance Questionnaire), and the PrEP Stigma Scale, with survey items tailored to evaluate PrEP acceptance, satisfaction, and perceptions of PrEP-related stigma for both the CAB-LA and oral PrEP arms.

## 4.2. Study Schema

Patients >18 y/o who are newly started on PrEP therapy at WVHR and have access to a smart phone with data (N=105)

- Participants will have been prescribed CAB-LA, daily FTC/TDF, or daily FTC/TAF in accordance with the WVHR standard of care by a licensed HCP prior to enrolling in the study
- II. Not receiving HIV PrEP care outside of WVHR
- III. No positive HIV diagnosis
- IV. No contraindications to oral or injectable PrEP therapy

# CAB-LA PrEP Arm n = 70

- PrEP injections at months0, 1, 3, 5, 7, 9 and 11
- Education modules at months 2, 4, 6, 8, and 10

# Oral PrEP Arm n = 35

- PrEP prescription fills at months0, 3, 6, 9, and 12
- Education modules at months 2,
  4, 6, 8, and 10

**Primary outcome measure:** Proportion of patients reporting persistence at months 3 and end of study, validated by medication possession ratio between the CAB-LA and Oral PrEP cohorts. Adherence assessed by estimating the proportion of participants who missed one or more injections or received injections outside the 7 day window and the proportion of participants who reported missing days of oral PrEP or with gaps > 90 days

**Secondary outcome measure 1**: retention in care in patients receiving CAB-LA vs oral PrEP defined as the proportion of patients presenting for their follow-up appointments within 30 days of their scheduled visit at months 3, 9 and 12 for the Oral PrEP cohort and at months 3, 9, and 11 for the CAB-LA cohort

**Secondary outcome measure 2:** patient-reported outcomes including PrEP medication satisfaction, PrEP acceptance, and PrEP-related stigma, and barriers to adherence and reasons for PrEP discontinuation assessed through brief behavioral surveys

**Secondary outcome measure 3**: implementation outcomes including patient acceptability (AIM), appropriateness (IAM), and helpfulness of the education modules within the digital health program assessed using a Likert scale and health literacy evaluation

**Secondary outcome measure 4:** clinician acceptability, appropriateness, and feasibility of implementing long-acting cabotegravir injections (AIM, IAM, FIM), and barriers to and facilitators for implementation of CAB-LA

#### 5. STUDY POPULATION

- 5.1. Inclusion Criteria
  - 5.1.1. >18 y/o
  - 5.1.2. Initiation of PrEP with CAB-LA, daily FTC/TDF, or daily FTC/TAF prescribed in accordance with the WVHR standard of care practices (based practices on CDC PrEP 2021 Clinical Practice Guidelines) by a licensed HCP
  - 5.1.3. PrEP dispensed by WVHR pharmacy
  - 5.1.4. Access to a smart phone
- 5.2. Exclusion Criteria
  - 5.2.1. <18 y/o
  - 5.2.2. Receiving HIV PrEP care outside of WVHR
  - 5.2.3. Positive HIV diagnosis
  - 5.2.4. Contraindication to oral or injectable PrEP therapy
  - 5.2.5. Receiving oral bridging therapy prior to injectable PrEP therapy
  - 5.2.6. Confirmed pregnancy
  - 5.2.7. Vulnerable populations
- 5.3. Study Sample
  - 5.3.1. n = 105 (70 CAB-LA intervention participants vs 35 oral PrEP participants)
- 5.4. Screening and Enrollment
  - 5.4.1. Patients will be enrolled on a rolling basis via HCPs at WVHR. HCPs will verify participant's eligibility for the study.

#### 6. STUDY INTERVENTIONS AND PROCEDURES

6.1. Study Procedures and Interventions Table (Figure 6a)

| CAB-LA PrEP Arm (N=70) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month 0 | Month 0 | Month 1 | Month 2 | Month 3 | Month 4 | Month 5 | Month 6 | Month 7 | Month 8 | Month 9 | Month 10 | Month 11 | Month 12 |
| Baseline labs<br>and<br>1st PrEP<br>injection<br>Baseline<br>demographic<br>survey | Baseline<br>evaluation<br>and<br>introduction<br>to support<br>group | 2nd PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>3rd PrEP<br>injection<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>4th PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>5th PrEP<br>injection<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>6th PrEP<br>injection<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>7th PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | PRO data<br>collection –<br>Set #2 |
| Oral PrEP Arm (N=35) | | | | | | | | | | | | | |
| Month 0 | Month 0 | Month 1 | Month 2 | Month 3 | Month 4 | Month 5 | Month 6 | Month 7 | Month 8 | Month 9 | Month 10 | Month 11 | Month 12 |
| Baseline labs<br>and<br>PrEP<br>prescription<br>filled<br>Baseline<br>demographic<br>survey | Baseline<br>evaluation<br>and<br>introduction<br>to support<br>group | Persistence<br>Assessment PRO data<br>collection –<br>Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Follow-up<br>labs and<br>PrEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Follow-up<br>labs and<br>PFEP<br>prescription<br>refill<br>Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Follow-up<br>labs and<br>PrEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Follow-up<br>labs and<br>PFEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment |
| Reciprocity App – Education Modules Month 2: PrEP Medicines Month 4:Protecting Yourself from HIV, STIs, and other infections Month 6: Building a Support System for HIV Prevention Month 8: Being an Active Participant in Your Own Care Month 10: Overcoming Stigma and Becoming a Health Advocate | | | PRO dat PrEP PrEP- | ence assess<br>a collectio<br>Medication S<br>Related Stig | n (Set #1):<br>Satisfaction | PRO da | | on (Set #2) | | | | | |

## 6.2. Description of Study Procedures

Before any screening procedure is performed, informed consent will be obtained. Labs will be taken at baseline and months 3, 5, 7, 9, and 11 for the CAB-LA cohort and at baseline and months 3, 6, 9, and 12 for the Oral PrEP cohort (only collected through standard of care). Participants will complete a baseline evaluation and be introduced to a support group at baseline. Patients will complete assessments within the TheraPay App. Clinicians will complete assessments outside of the app. Patients in both cohorts will complete baseline demographic surveys in month 0, patient reported outcomes (PRO) data collection set 1 in months 1, 5, and 11 and PRO data collection set 2 in months 3, 9, and 12. Patients in the CAB-LA PrEP cohort will complete persistence assessments in months 1, 3, 5, 7, 9, and 11. Patients in the Oral PrEP cohort will complete persistence assessments every month from months 1 through 12. Clinic staff will complete surveys at baseline, month 6, month 12, and at the end of the study. The

schedule of assessments for the CAB-LA PrEP cohort, Oral PrEP cohort, and clinicians is presented in figure 6a. Instruments are in Appendix B for the CAB-LA cohort, in Appendix C for the Oral PrEP cohort, and Appendix D for clinicians. Patient incentives for completing the assessment activities are outlined in Appendix E.

- 6.2.1. Baseline Patient Demographic Survey
- 6.2.2. Medication Persistence
  - 6.2.2.1. Definition: Continue to take medicines over time independent of adherence to the PrEP medication regimen.
- 6.2.3. Persistence Assessment CAB-LA
  - 6.2.3.1. The proportion of participants who received at least one PrEP injection who remained on injectable PrEP or oral bridging at months 3 and 11 measured by the self-report assessment and validated with claims data.
- 6.2.4. Persistence Assessment Oral PrEP
  - 6.2.4.1. The proportion of participants who initiated oral PrEP who remained on oral PrEP at months 3 and 12 measured by the self-report assessment and validated with claims data period.
- 6.2.5. Adherence
  - 6.2.5.1. Definition: Taking PrEP in line with medical advice/using PrEP appropriately (critical for efficacy).
- 6.2.6. Adherence Assessment CAB-LA
  - 6.2.6.1. Adherence to the dosing schedule will be assessed at month 3 (early adherence) and end of study by:
    - A) Estimating the number of individuals who missed one or more consecutive injections without taking daily oral bridging PrEP while not on CAB-LA injections and mean and median number of injections missed during a 6- and a 12-month period.
- 6.2.7. B) Estimating the number of individuals who received the injections seven or more days later than their scheduled injection visit and the mean and median duration of delayed injections. Adherence Assessment Oral PrEP

- 6.2.7.1. Adherence to the dosing schedule will be assessed at months 3 (early adherence) and 12 by:
  - A) Estimating the number of individuals who reported three or more days of oral PrEP missed and the mean and median number of days they missed.
  - B) Estimating the number of individuals who had a gap of >90 days between the end of the days of supply of a dispensing and the start date of the next fill.

## 6.2.8. Patient Reported Outcomes

- 6.2.8.1. Patient Reported Outcomes Set 1: PrEP Medication Satisfaction, PrEP-Related Stigma, Acceptability of Intervention Measure (AIM)
- 6.2.8.2. Patient Reported Outcomes Set 2: PrEP Acceptance, Intervention Appropriateness Measure (IAM)
- 6.2.8.3. Helpfulness of the education modules and Health Literacy Evaluation

#### 6.2.9. Clinician Instruments

## 6.2.9.1. Baseline Provider Survey

- 6.2.9.1.1. Information About You and Your Patients
- 6.2.9.1.2. Acceptability of Intervention Measure (AIM)
- 6.2.9.1.3. Intervention Appropriateness Measure (IAM)
- 6.2.9.1.4. Feasibility of Intervention Measure (FIM)
- 6.2.9.1.5. Barriers and Facilitators for Implementation of Long-Acting

  Cabotegravir for PrEP

### 6.2.9.2. Follow-up Provider Survey

- 6.2.9.2.1. Information About You and Your Patients
- 6.2.9.2.2. Acceptability of Intervention Measure (AIM)
- 6.2.9.2.3. Intervention Appropriateness Measure (IAM)
- 6.2.9.2.4. Feasibility of Intervention Measure (FIM)
- 6.2.9.2.5. Barriers and Facilitators for Implementation of Long-Acting

  Cabotegravir for PrEP

#### 6.3. Standard of Care Visits

- 6.3.1. The standard of care for patient visits will not be affected. The patients will only be given additional surveys to complete.
- 6.4. Follow-Up Visits
  - 6.4.1. CAB-LA PrEP cohort: 2<sup>nd</sup> PrEP injection at month 1; follow-up labs and PrEP injections in months 3, 5, 7, 9, and 11.
  - 6.4.2. Oral PrEP cohort: follow-up labs and prescription refills in months 3, 6, 9, and 12.
- 6.5. Switching between PrEP regimens
  - 6.5.1. To be included in final data analysis, participants cannot switch between PrEP regimens before 6-months duration of initial PrEP.
- 6.6. PrEP Discontinuation
  - 6.6.1. Participants will be deemed as having discontinued PrEP if they miss more than 3 consecutive months for PrEP.
  - 6.6.2. Participants will be called, texted and emailed for three consecutive months before considered them as discontinued.
- 6.7. STI Screening and Management
  - 6.7.1. Participants will receive STI screening at baseline and at every follow up clinic visit.

    Participants will be screened if they present with any type of symptoms that

    warrant STI testing. If a participant tests positive for an STI other than HIV, they will

    receive guideline-directed therapy at the discretion of their HCP at WVHR.
- 6.8. Suspected or Confirmed HIV Infection
  - 6.8.1. HIV screening will occur a minimum as recommended for every 2 months with CAB-LA (same time as injections) and every 3 months for oral PrEP.
- 6.9. PrEP Choice Counselling
  - 6.9.1. Patients will be counseled on the benefits and risks of both oral PrEP and PrEP injections. The selection of PrEP option will be done as the standard of care through shared-decision with the patient.
- 6.10. Possible Participant Pathways

6.10.1. There will only be two observational cohort arms. Patients will either be placed into the injectable PrEP arm or the oral PrEP arm based on their baseline prescription.

### 6.11. Adherence Strategies

- 6.11.1. Patients on oral PrEP will be encouraged to set a daily reminder on their smart phone as an alarm at the time their dose is due.
- 6.11.2. Patients on injectable PrEP will set a monthly calendar reminder on the day/time their injection is due.

#### 6.12. Retention Strategies

- 6.12.1. Follow-up appointments will be set up and conveyed at each appointment.
- 6.12.2. Reminder calls will be made by a staff member a few days before the appointment.
- 6.13. Interventions: PrEP Initiation and Digital Health Companion Program
  - 6.13.1. Participants will be enrolled in the CAB-LA and Oral PrEP cohorts. Participants in the CAB-LA cohort will receive their first dose of the PrEP injection at month 0.

    Injections will also be administered in months 1, 3, 5, 7, 9, and 11. Participants in the Oral PrEP cohort will have their prescription filled at month 0, 3, 6, 9, and 12.

    The schedule of dosing is presented in Figure 6a.
  - 6.13.2. Participants in both cohorts will complete education modules and health literacy evaluations in the TheraPay App in months 2, 4, 6, 8, and 10 as presented in Figure 6a. Education Modules include PrEP Medicines (month 2), Protecting Yourself from HIV, STIs, and other infections (month 4), Building a Support System for HIV Prevention Month 6: Being an Active Participant in Your Own Care (month 8), and Overcoming Stigma and Becoming a Health Advocate (month 10).

#### 6.14. STATISTICAL ANALYSIS

- 6.14.1. Study Endpoints
  - 6.14.1.1. Medication Adherence and PersistenceMedication persistence is defined as continuing to take PrEP over timeindependent of adherence to the medication regimen. The proportion of

patients reporting receipt of CAB-LA or oral PrEP at months 3 (early) and end of study (late) will be measured through patient questionnaires and validation protocols. Medication adherence is defined as taking PrEP in line with medical advice.

#### 6.14.1.2. Retention-in-Care

Retention-in-care is defined as the proportion of patients presenting for their follow-up appointments within 30 days of their scheduled visit at months 3, 9, and 12 after PrEP initiation in the oral PrEP cohort and months 3, 9, and 11 for the CAB-LA cohort.

## 6.14.1.3. Patient-reported Outcomes

Patient-reported outcomes will be assessed through surveys. Medication satisfaction will be measured by the HIV Treatment Satisfaction Questionnaire (HIVSTQ) adapted for PrEP and PrEP stigma will be measured by the PrEP Stigma Scale at months 1, 5, and 11. PrEP acceptance will be measured by the Modified Injection Treatment Acceptance Questionnaire (Modified I-TAQ) at months 3, 9, and 12. Barriers to adherence to oral PrEP and reasons for PrEP discontinuation will be assessed through brief behavioral surveys every month after the initiation of PrEP. Barriers to adherence to CAB-LA injections and reasons for PrEP discontinuation will be assessed through brief behavioral surveys at months 1, 3, 5, 7, 9, and 11.

## 6.14.1.4. Implementation Outcomes for the Mobile App

Acceptability of the mobile app to support patients in taking PrEP will be measured by the Acceptability of Intervention Measure (AIM) at months 1, 5, and 11. Appropriateness of the mobile app to support patients in taking PrEP will be measured by the Intervention Appropriateness Measure (IAM) at months 3, 9, and 12.

6.14.1.5. Clinic Staff Acceptability, Appropriateness, and Feasibility of Providing Long-acting Cabotegravir Injections

Acceptability of the process for providing long-acting cabotegravir injections will be assessed by the Acceptability of Intervention Measure (AIM). Appropriateness of the process for providing long-acting cabotegravir injections will be assessed by the Intervention Appropriateness Measure (IAM). Feasibility of long-term use of cabotegravir injections will be assessed by the Feasibility of Intervention Measure (FIM). Willingness to sustain provision of long-acting cabotegravir injections and barriers to and facilitators for provision of long-acting cabotegravir injections will be assessed through a brief survey. The clinic staff surveys will be administered at baseline, month 6, month 12, and end of study.

## 7. Statistical Analyses

Baseline analyses will include tabulations of demographic and clinical variables of the study participants. Chi-square tests and t-tests will be used to compare these groups to determine if baseline differences exist. The distribution of each continuous variable will be inspected for outliers to determine whether a parametric or non-parametric approach should be applied. The Wilcoxon ranked sum test will be used for any variable that does not meet the statistical assumptions of the t-test. Variables found to be associated with persistence or adherence following univariate analysis will be included in multivariate models.

To assess the co-primary endpoint of persistence at 3 months and end of study, the proportion of participants reporting continued receipt of injections in the CAB-LA cohort and the proportion of patients reporting continued use of PrEP by mouth in the oral PrEP cohort on the persistence assessment will be compared using chi square tests or Fisher's exact tests. Self-reported persistence will be validated by the medication possession ratio (MPR). MPR is defined as the number of days of medication dispensed during the study period divided by the number of days that the person should have received therapy. The percent of CAB-LA participants with MPRs  $\geq$  1.0 will be compared to the percent of oral PrEP participants with MPRs  $\geq$  1.0 using chi square tests or Fisher's exact tests. To assess the co-primary endpoint of adherence, chi square tests or Fisher's

exact tests will be used to compare the percent of CAB-LA participants who reported missing one or more injections during the study period to the percent of oral PrEP participants who reported three or more missed days of oral PrEP. The percent of CAB-LA participants who received any injections seven or more days later than their scheduled injection or oral PrEP participants who had a gap of >90 days between the end of the days of supply of a dispensing and the start date of the next fill will be compared.

## Sample Size

Assuming adherence proportions of .90 and .65 and sample sizes of 70 and 35 in the CAB-LA and oral PrEP arms respectively, the 95% confidence interval for the difference between the CAB-LA proportion and the oral PrEP proportion is .0771 to .4229.

#### 8. SAFETY MONITORING AND ADVERSE EVENT REPORTING

- 8.1. An adverse event (AE) is defined as any untoward medical occurrence whether thought to have been caused by the investigational medical product or the Study or not, and a Serious Adverse Event (SAE) shall mean any adverse event which is fatal, life threatening, disabling or incapacitating, requires in-patient treatment or prolongs existing hospitalization, is a congenital anomaly in the off-spring of the patient or which may require intervention to prevent the previously stated outcomes.
- 8.2. All AEs should be reported via FEARS by the health care providers. All SAEs and medical device incidents considered related to CAB-LA should be reported to GSK within 24 hours of awareness. All pregnancies associated with CAB-LA (initial notification followed by outcome of the mother and infant) should be reported to GSK within 1 week of awareness.
- 8.3. Participants will be counselled by HCPs at WVHR on the common ADEs to be aware of and when the participants should contact their HCP. Common ADEs can also be found in the FDA package insert. Participants will be counselled that If they become pregnant or suspect they might be pregnant, they should contact their HCP. All investigators and health care providers are strongly encouraged to report all pregnancies exposed to Cabotegravir to the Antiretroviral Pregnancy Registry (APR) as soon as the pregnancy is

identified. Pregnancies can be reported to the Registry at SM\_APR@APRegistry.com via the data forms available at www.APRegistry.com

#### 9. HUMAN PARTICIPANTS AND DATA PROTECTION

### 9.1. TheraPay App

9.1.1. The TheraPay requires a username and password to access the program and data stored by the application. Only survey completed by enrolled participants will be stored within the application along with name, phone number, and email address.

#### 10. TIMELINES

10.1. Patients will be enrolled until the n value of 105 is met.

| 2-3 months | 3-6 months* | 12 months | 3 months |
|---|---|---|---|
| Development of study protocol, | Participant enrollment | Study period | Data analysis and |
| educational modules and survey | (rolling basis) | | publication |
| instruments | | | submission |

#### 11. PRESENTATION AND PUBLICATION PLANS

#### 12. REFERENCES

- 12.1. Huang YLA, Tao G, Smith DK, Hoover KW. Persistence with Human Immunodeficiency Virus Pre-exposure Prophylaxis in the United States, 2012-2017. Clin Infect Dis. 2021;72(3):379-385.
- 12.2. Keyes J, Crouse EC, DeJesus E, Rolle C-P. Determinants of pre-exposure prophylaxis (PrEP) persistence in a high-risk population in Central Florida. J Investig Med. 2021;69(2):397 LP 401.
- 12.3. Spinelli MA, Scott HM, Vittinghoff E, et al. Missed Visits Associated with Future Preexposure Prophylaxis (PrEP) Discontinuation among PrEP Users in a Municipal Primary Care Health Network. Open Forum Infect Dis. 2019;6(4).
- 12.4. Krakower D, Maloney KM, Powell VE, et al. Patterns and clinical consequences of discontinuing HIV preexposure prophylaxis during primary care. J Int AIDS Soc. 2019;22(2):1-9.
- 12.5. Czarnogorski M, Garris C, D'Amico R, et al. CUSTOMIZE: overall results from a hybrid III implementation-effectiveness study examining implementation of cabotegravir and

- rilpivirine long-acting injectable for HIV treatment in US healthcare settings; final patient and provider data. In: International AIDS Society Conferences on HIV Science.; 2021.
- 12.6. Garris C, Stassek L, D'Amico R, et al. Qualitative Patient-Participant Perspectives on Implementation of Monthly Cabotegravir and Ripilvirine Long-Acting (CAB+RPV LA) Injectable in the United States (CUSTOMIZE). IDWeek 2021. Abstract 883.
- 12.7. West Virginia Bureau for Medical Services. Preferred Drug List and Coverage Detail.s.

  Available at <a href="https://dhhr.wv.gov/bms/BMS Pharmacy/pages/preferred-drug-list.aspx.">https://dhhr.wv.gov/bms/BMS Pharmacy/pages/preferred-drug-list.aspx.</a>

  Accessed 09/06/2022.
- 12.8. Centers for Disease Control and Prevention. Vulnerable Counties and Jurisdictions Experiencing or At-Risk of Outbreaks. Available at https://www.cdc.gov/pwid/vulnerable-counties-data.html. Accessed 09/06/2022.
- 12.9. Centers for Disease Control and Prevention. HIV in the United States and Dependent Areas. Available at https://www.cdc.gov/hiv/statistics/overview/ataglance.html. Accessed 09/06/2022.
- 12.10. Schneider KE, White RH, O'Rourke A, et al. Awareness of and Interest in Oral Pre-Exposure Prophylaxis (PrEP) for HIV Prevention and Interest in Hypothetical Forms of PrEP among People who Inject Drugs in Rural West Virginia. AIDS Care. 2021;33(6):721-728.
- 12.11. Weitzman PF, Zhou Y, Kogelman L, Rodarte S, Vicente SR, Levkoff SE. MHealth for pre-exposure prophylaxis adherence by young adult men who have sex with men. mHealth. 2021;7(6).
- 12.12. Garrison LE, Haberer JE. Pre-exposure Prophylaxis Uptake, Adherence, and Persistence: A Narrative Review of Interventions in the U.S. Am J Prev Med. 2021;61(5 Suppl 1):S73-S86.
- 12.13. Deloitte. Medicaid and Digital Health: Findings from the Deloitte 2018 Survey of US Health Care Consumers. Available at <a href="https://www2.deloitte.com/us/en/insights/industry/public-sector/mobile-health-care-app-features-for-patients.html">https://www2.deloitte.com/us/en/insights/industry/public-sector/mobile-health-care-app-features-for-patients.html</a>. Accessed 09/06/2022.

- 12.14. Woodcock A, Bradley C. Validation of the HIV treatment satisfaction questionnaire (HIVTSQ). Qual life Res an Int J Qual life Asp Treat care Rehabil. 2001;10(6):517-531.
- 12.15. Arnould B, Gilet H, Patrick DL, Acquadro C. Item Reduction, Scoring, and First Validation of the ACCEPTance by the Patients of their Treatment (ACCEPT©)

  Questionnaire. Patient. 2017;10(1):81-92.
- 12.16. Klein H, Washington TA. The Pre-Exposure Prophylaxis (PrEP) Stigma Scale: Preliminary findings from a pilot study. Int public Heal J. 2019;11(2):185-195.
- 12.17. Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017;12(1):1-12.
- 12.18. Reciprocity Health. Available at https://www.reciprocityhealth.com/. Accessed 09/06/2022.
- 12.19. Fallon S, Molnar K, Taneva E, Simone L, Carter J, Sapir T. Tackling the HIV Epidemic in South Florida: Patient Insights on Approaches for HIV Counseling, Testing, and Access to Prevention or Treatment. Poster presentation at ID Week iNNOVATE RFP CAB LA for PrEP. October 21-25, 2020.
- 12.20. Felzien G, McIntosh S, Taneva E, et al. Do Patients and Healthcare Professionals See Eye-to-Eye on the Usefulness of Strategies for Promoting HIV Care? Poster presentation at ID Week. Washington, DC; October 2–6, 2019.
- 12.21. Taneva E, Simone L, Carter J, Sapir T, Brinson C, Wohl D. Taneva E, Simone L,
  Carter J, Sapir T, Brinson C, Wohl DA. Impact of Quality-Driven Interventions and Action
  Plans on Retention-in-care in 11 HIV Clinics. Poster presentation at the American
  Conference for the Treatment of HIV (ACTHIV). Miami, FL; April 1.
- 12.22. Wohl D, Brinson C, Hicks C, et al. Real-World Insights into Quality Improvement across 11 HIV Clinics in the US. Presentation at ID Week 2018. San Francisco, CA; October 3-7, 2018.
- 12.23. Glasgow RE, Harden SM, Gaglio B, et al. RE-AIM planning and evaluation framework: Adapting to new science and practice with a 20-year review. Front Public Heal. 2019;7(MAR).

12.24. Proctor E, Silmere H, Raghavan R, et al. Outcomes for implementation research:

Conceptual distinctions, measurement challenges, and research agenda. Adm Policy

Ment Heal Ment Heal Serv Res. 2011;38(2):65-76.

#### 13. APPENDICES

- 13.1.1. Informed Consent
- 13.1.2. CAB-LA PrEP ARM Instruments
  - 13.1.2.1. Baseline Demographic Survey
  - 13.1.2.2. Persistence Assessment
  - 13.1.2.3. Patient Reported Outcomes Set 1: PrEP Medication Satisfaction, PrEP-Related Stigma, Acceptability of Intervention Measure (AIM)
  - 13.1.2.4. Patient Reported Outcomes Set 2: PrEP Acceptance, Intervention Appropriateness Measure (IAM)
  - 13.1.2.5. Health Literacy Evaluations
- 13.1.3. Oral PrEP ARM Instruments
  - 13.1.3.1. Baseline Demographic Survey
  - 13.1.3.2. Persistence Assessment
  - 13.1.3.3. Patient Reported Outcomes Set 1: PrEP Medication Satisfaction, PrEP-Related Stigma, Acceptability of Intervention Measure (AIM)
  - 13.1.3.4. Patient Reported Outcomes Set 2: PrEP Acceptance, Intervention Appropriateness Measure (IAM)
  - 13.1.3.5. Health Literacy Evaluations
- 13.1.4. Clinician Instruments
  - 13.1.4.1. Baseline Provider Survey
  - 13.1.4.2. Acceptability of Intervention Measure (AIM)
  - 13.1.4.3. Intervention Appropriateness Measure (IAM)
  - 13.1.4.4. Feasibility of Intervention Measure (FIM)
  - 13.1.4.5. Follow-up Provider Survey
- 13.1.5. Incentive Mapping
- 13.1.6. List of Tables
  - 13.1.6.1. Study Procedures
- 13.1.7. List of Figures
  - 13.1.7.1. Study Schema

## 13.1.7.2. Study Timelines

13.1.8. Forms for Safety Reporting

## 1. PROTOCOL SUMMARY

| Title | A Transformative Approach Utilizing Behavioral Economics, Education, |
|---|---|
| | and Data Science to Support Patients Initiating PrEP with Retention-in- |
| | care and Medication Persistence |
| Funder | ViiV Healthcare |
| Study Design | Observational Cohort Study |
| Study Population | Patients >18 y/o who are newly started on PrEP at WVHR and have |
| | access to a smart phone with data. |
| Study Size | n = 105 (70 CAB-LA intervention participants and |
| | 35 oral PrEP participants) |
| Study Duration | 12 months |
| Study Site(s) | West Virginia Health Right |
| Intervention | Participants will have been prescribed CAB-LA, daily FTC/TDF, or daily |
| Description | FTC/TAF in accordance with the WVHR standard of care by a licensed |
| | HCP prior to enrolling in the study. Those receiving CAB-LA will be in |
| | one arm and those receiving oral therapy will be in the other arm of |
| | the study. |
| Study Aim | To determine the persistence in injectable PrEP compared to Oral |
| | PrEP therapy |
| Primary Objectives | To evaluate medication persistence in patients receiving CAB-LA |
| | vs oral PrEP and who engage with a digital health companion |
| | program |
| Secondary | Evaluate Retention-in-care in patients receiving CAB-LA vs oral |
| Objective 1 | PrEP |
| Secondary | Evaluate PROs (including PrEP medication satisfaction, PrEP |
| Objective 2 | acceptance, stigma, and reasons for PrEP discontinuation) in |
| | patients receiving CAB-LA vs oral PrEP |
| Secondary | Evaluate the acceptability, appropriateness, and helpfulness of a |
| Objective 3 | digital health companion program for PrEP |

| Secondary | Evaluate the acceptability, barriers to, and facilitators for |
|-------------|---------------------------------------------------------------|
| Objective 4 | implementation of CAB-LA |

## Study Schema Figure

Figure showing study components and flow – organize by participant cohort (i.e. oral, LA, no PrEP)

## Study Outcomes Table

| Primary or Secondary | Definitions | Type of | Assessment | Data Source | Intervention | Tool/Instrument |
|---|---|---|---|---|---|---|
| Endpoint | | Endpoint | Timepoint | | or Approach | for Endpoint |
| 1. Primary Endpoint: PrEP | Proportion of patients | Quantitative | M3 and end | Participant survey | Participant | Survey and |
| adherence and Persistence | reporting receipt of CAB- | | of study | and EHR | survey and EHR | Medication |
| | LA injections or use of | | | | | Retention Ratio |
| | oral PrEP at 3 months | | | | | |
| | after PrEP initiation and | | | | | |
| | end of study | | | | | |
| 2. Secondary Endpoint: | The proportion of | Quantitative | M3, M9, | Participant survey | Participant | Survey |
| Retention-in-care | patients presenting for | | M11, M12 | and EHR | survey and EHR | |
| | their follow-up | | | | | |
| | appointments within 30 | | | | | |
| | days of their scheduled | | | | | |
| | visit at months 3, 9 and | | | | | |
| | 12 after PrEP initiation | | | | | |
| | for the Oral PrEP arm | | | | | |
| | and months 3, 9, and 11 | | | | | |
| | for the CAB-LA arm. | | | | | |
| 3. Secondary Endpoint: PROs | PRO Set #1: | Qualitative | M1, M5, M11 | Participant Survey | Patient | Survey |
| | PrEP Medication | | (PRO Set #1), | | questionnaire | |
| | Satisfaction; PrEP- | | | | | |
| | Related Stigma | | M3, M9, M12 | | | |
| | | | (PRO Set #2) | | | |
| | PRO Set #2: PrEP | | | | | |
| | Acceptance | | Barriers to | | | |
| | | | adherence in | | | |
| | Barriers to adherence to | | oral PrEP | | | |
| | CAB-LA injections and | | arm: M1, M2, | | | |
| | | | M3, M4, M5, | | | |

| | oral PrEP, and reasons | | M6, M7, M8, | | | |
|---|---|---|---|---|---|---|
| | for PrEP | | M9, M10, | | | |
| | discontinuation will be | | M11, M12 | | | |
| | assessed through brief | | | | | |
| | behavioral surveys | | Barriers to | | | |
| | | | adherence in | | | |
| | | | CAB-LA PrEP | | | |
| | | | arm: M1, M3, | | | |
| | | | M5, M7, M9, | | | |
| | | | M11 | | | |
| 4. Secondary Endpoint: | Acceptability of | Qualitative | M3, M9, M12 | Participant Survey | Patient | Survey |
| Implementation Outcomes | Intervention Measure | | | | questionnaire | |
| | (AIM) and Intervention | | | | | |
| | Appropriateness | | | | | |
| | Measure (IAM) | | | | | |
| | Health literacy | | | | | |
| | evaluation and | | | | | |
| | helpfulness of the | | | | | |
| | education modules | | | | | |
| | within the digital health | | | | | |
| | program assessed | | | | | |
| | through a brief survey | | | | | |
| 5. Secondary Endpoint: | Acceptability of | Qualitative | M0, M6, | Clinician Survey, | Clinician Survey, | Clinician Survey, |
| Clinician Acceptability, | Intervention Measure | | M12, and End | Interview | Interview | Interview |
| Appropriateness, and | (AIM), Intervention | | of Study | | | |
| Feasibility | Appropriateness | | | | | |
| | Measure (IAM), and | | | | | |
| | Feasibility of | | | | | |
| | Intervention Measure | | | | | |
| | (FIM) | | | | | |

| Willingness to sustain |
|--------------------------|
| provision of CAB-LA, |
| barriers to and |
| facilitators for |
| provision of CAB-LA |
| assessed through a brief |
| survey |

## Appendix A: Informed Consent

#### **SUMMARY**

We are asking you to be in a research study to determine the helpfulness of using a cell phone application in supporting patients wanting to participate in HIV prevention care. TheraPay Rewards is a mobile and web program that tracks the care and rewards patients for doing activities such participating in education activities and completing surveys about their care. The app provides information on what activities the patient needs to do to earn rewards. It also sends reminders along the way. This will help us understand if the overall patient experience and satisfaction improves when compared to the traditional care and education approaches. This form explains what you need to know to decide whether you want to participate in this program

## What will I be expected to do in this study?

You will have to download the TheraPay app. Also, consent to us telling notifying you of when education and surveys will be available for you to complete. In order to receive rewards you would be required to complete the education and surveys during the specified times that they are designated to be completed.

## Are there any risks to being in the study?

There is minimal risk. The level of risk you might experience in everyday life, is associated with this study. The risks primarily reside in your personal information being compromised. Payment occurs in the form of rewards added to a reloadable smart rewards card from TheraPay. This reward card will be sent in the mail to you.

Side effects associated with PrEP are possible. To find further information about possible side effects, read the drug label or package insert or talk to your health care provider. If you experience side effects associated with PrEP, contact your healthcare provider. If you become pregnant or suspect that you might be pregnant, contact your healthcare provider.

## Will I benefit from being in the study?

You will not benefit directly from the study. We hope to learn how to best communicate and support patients with HIV prevention care activities for patients in the future.

### Will my study information be kept safe?

Yes. All your health information is kept private and not shared with anyone. To learn more, go online to: TheraPay's Privacy Policy at <a href="https://www.therapayrewards.com/privacy-policy">www.therapayrewards.com/privacy-policy</a>. The Therapay app will not connect with your contacts or social media.

#### Is there any cost for me from being in this study?

There is no cost to you for being in the study. You will be responsible for the cost of your regular care. Additionally, there may be costs for data usage relating to the TheraPay application.

## Will I get any money or gifts for being in this study?

Participants will be rewarded for completing tasks assigned to them while receiving care for HIV prevention. You will receive your rewards card (similar to a debit card) in the mail in 1 to 2 weeks after registering for TheraPay. You will get information about the activities and rewards you qualify for via the TheraPay Rewards app, emails, and text messages. A \$5-30 credit per task will be issued to your gift card. You will need to complete approximately 20-25 tasks over 12-months. A maximum of \$265 will be loaded onto the card.

### Other information

Your information collected as part of this research will not be share with without unique identifiers being removed. You can contact Rhonda Francis, 304-414-5922 if you have questions about this study.

### **Giving consent**

We will ask you to sign this document. By signing this document, you are agreeing participation in this study. Make sure you understand what the study is about before you sign.

#### HIPAA Authorization - For the Use of Patient Information for Research

The purpose of this section of the form is to give your permission to the research team to obtain and use your Protected Health Information (PHI) or patient information. Your patient information will be used to do the research described earlier in this form. State and federal privacy laws protect your patient information. These laws say that, in most cases, your health care provider can release your identifiable patient information to the research team only if you give permission by signing this form.

You do not have to sign this form. If you do not, you will not be allowed to join the research study. Your decision to not sign this form will not affect any other treatment, health care, enrollment in health plans or eligibility for benefits.

"Patient information" means the health information in your medical or other healthcare records. It also includes information in your records that can identify you. For example, it can include your name, address, phone number, birthdate, and medical record number.

By signing this form, you are giving permission to the following organization(s) to disclose your patient information for this research.

- West Virginia Health Right
- Reciprocity Health, Inc.

Patient information that will be released for research use This permission is for the health care provided to you during the following time period: From the time of enrollment for a duration of approximately 12-months.

The information that will be released and used for this research is described below:

- First Name (You will share this with the app)
- Last Name (You will share this with the app)

- DOB (You will share this with the app)
- Email (You will share this with the app)
- Mobile Number (You will share this with the app)
- Gender (You will share this with the app)
- Address (You will share this with the app)
- Confirmation of tasks (You will share this with the app)
- HIV Prevention Care Information (Will be shared)

## How your patient information will be used?

## 1. Who may get your patient information?

• The group funding the study, known as the sponsor of this research. "Sponsor" includes any persons or companies that are working with or for the sponsor, or that are owned by the sponsor

## 2. Why your patient information will be used and/or given to others

- To do the research
- To study the results, and
- To see if the research was done right

If the results of this study are made public, information that identifies you will not be used. The researcher will use your patient information only in the ways that are described in this research consent form and this HIPAA Authorization. You can ask questions about what the research team will do with your information and how they will protect it.

The privacy laws do not always require the people who get your information to keep your information confidential. After your information has been given to others, there is a risk that it could be shared without your permission. This permission for the researchers to obtain your patient information ends when the research ends and any required monitoring of the study is finished.

## **Canceling your permission**

You may change your mind at any time. To take back your permission, you must send your written request to:

Rhonda Francis WV Health Right 1520 East Washington Street Charleston, WV 25311 Phone: 304-414-5922

If you take back your permission, the research team may still keep and use any patient information about you that they already have. But they can't obtain more health information

about you for this research unless it is required by a federal agency that is monitoring the research.

If you take back your permission, you will need to leave the research study. This means that you would not have any more notifications or rewards. Changing your mind will not affect any other treatment, payment, health care, enrollment in health plans or eligibility for benefits.

## **Giving permission**

By signing this document, you are agreeing to participation in this study. You are also agreeing that your patient information will be used as we described earlier in this form. We will give you a copy of this document for your records. We will keep a copy with the study records.

If you have any questions about the study after you sign this document, you can contact the study team using the information provided above. I have read this consent and HIPAA Authorization form describing the research study and how my patient information will be used. I have had a chance to ask questions and I have received answers to my questions. I agree to be in this study. I also agree to the use of my patient information for this research.

| Printed Name of Research Subject |
|---------------------------------------------------------|
| Signature of Decearch Subject Date of signature |
| Signature of Research Subject Date of signature |
| Printed Name of Person Obtaining Consent |
| Signature of Person Obtaining Consent Date of signature |

# PrEP Digital Health Companion Clinician Survey Informational Sheet

**Introduction:** You are being invited to volunteer for a research study. You must read each item in this before you agree to take part in this study. This form will give you more information about this study. You should not continue with the survey if you have questions after reading the information sheet.

**Purpose of the research:** The intent of this study is to gather valuable insights on unmet needs and challenges in PrEP and to gauge Health Care Provider's (HCP's) views on potential solutions for overcoming specific barriers such utilization of a digital health companion. From the information collected and studied, we plan to learn more about the quality of care for patients HIV prevention needs. About 10 clinicians will complete this survey.

What you will do in this research: You are being asked to volunteer as a participant for a short survey. The survey will take approximately 5-10 minutes. You will complete one survey intended to obtain your viewpoint about the healthcare experiences of your patients with influenza.

**Risks:** There are no foreseeable risks for you because the information being collected will not be linked back to your name or your specific patients.

**Benefits:** Your answers to questions will help inform future clinical education for providers in HIV prevention care. You will receive a de-identified summary report of aggregate responses through a live virtual continuation education presentation. The de-identified data collected for this project may be published in a peer-reviewed manuscript or presented in a national conference to inform other providers the barriers in care for patients.

Compensation: A \$50 gift card will be offered for completion of this survey

**Confidentiality:** Your responses will be kept confidential. When research results are reported, responses will be deidentified and aggregated.

**Participation and withdrawal:** Your participation in this survey is completely voluntary. You may refuse to participate, which will disenroll. At any time during the survey you exit and cease your participation. However, once answers have been submitted, they cannot be retracted as the data is deidentified.

**To Contact the Researcher:** If you have questions or concerns about this research, please contact: Dr. Jeff Carter: Phone: 954-718-6055 ext 23; Address: 114 5th Ave, 14th Floor New York, NY 10011 Email: j.carter@primeinc.org.

By continuing to complete the online survey form you are consenting to participate in the survey.

Please save a copy of this communication for your records.

Appendix B: CAB-LA PrEP Arm Instruments

**<u>Activity Title</u>**: Baseline Information About You

<u>Activity Description:</u> Today we'll ask you to answer some questions about yourself. The survey is 17 questions and should take about 10 minutes to complete.

## **Baseline Demographic Survey**

| Question | Question |
|---|---|
| | # |
| What year were you born? [Write in] | 1 |
| Which of the following best describes your racial/ethnic background? (Select all that apply) | |
| ☐ African American/Black | |
| ☐ Asian/Pacific Islander | |
| ☐ Caucasian/White | 2 |
| ☐ Hispanic/Latinx | |
| ☐ Native American/Alaska Native | |
| ☐ A race or ethnicity not listed: [Write in] | |
| How do you describe your gender? (Select 1) | |
| □ Female | |
| □ Male | |
| ☐ Transgender woman | 3 |
| ☐ Transgender man | |
| □ Non-binary | |
| ☐ A gender not listed: [Write in] | |
| How do you describe your sexual orientation? (Select 1) | |
| ☐ Heterosexual/Straight | |
| ☐ Gay or Lesbian | |
| ☐ Bisexual | 4 |
| ☐ Queer or Sexually Fluid | |
| □ Pansexual | |
| ☐ A sexual orientation not listed: [Write in] | |
| What is the highest degree or school level you have completed? (Select 1) | |
| ☐ Primary school | |
| ☐ Some high school | |
| ☐ High school diploma or GED | |
| ☐ Some college | 5 |
| □ 2-year college degree | |
| ☐ 4-year college degree | |
| ☐ Graduate level degree | |
| ☐ A school level not listed: [Write in] | |
| What health coverage are you currently enrolled with? (Select up to 2) | |
| □ Medicaid | 6 |
| ☐ Medicare | 0 |
| ☐ Affordable Care Act | |

| | Uninsured | |
|---|---|---|
| | Private health insurance | |
| | A health coverage not listed: [Write in] | |
| Why ar | e you using pre-exposure prophylaxis (PrEP) to prevent HIV? [Select all that apply] | |
| | Reduce acquisition of HIV from sex | 7 |
| | Reduce acquisition of HIV from IV drug use | |
| The | next 5 questions ask about your food, housing, and transportation routines from the | past 12 |
| montl | hs. If you have concerns and need support, please check in with your provider at you | r next visit |
| | or call 2-1-1 for immediate support. | |
| | ast 12 months, was there a time when you were not able to pay the mortgage or | |
| rent on | | |
| | No<br> | 8 |
| | Yes | |
| <u> </u> | Not applicable | |
| | ast 12 months, was there a time when you did not have a steady place to sleep or | |
| siept in | a shelter (including now)? | 9 |
| | No<br> | |
| <u> </u> | Yes | |
| | ast 12 months, have you or the people you live with been unable to get utilities | |
| (neat, e | electricity) when it was really needed? | 10 |
| | No | |
| \ | Yes | |
| | the past 12 months, the food you bought just didn't last and you didn't have money | |
| to get r | | 4.4 |
| | Never true | 11 |
| | Sometimes true | |
| \ | Often true | |
| | the past 12 months, has lack of transportation kept you from medical appointments, | |
| _ | your medicines, non-medical meetings or appointments, work, or from getting | 12 |
| unings u | that you need? | 12 |
| | No<br>Yos | |
| Do you | Yes feel physically and emotionally safe where you currently live? | |
| | Yes | 13 |
| | No | 13 |
| During | the past 30 days, have you used any of the following? | |
| During | An illegal drug (such as by snorting it or injecting it) | |
| • | Pain killer to get high (like OxyContin, sometimes called Oxy or OC) or Percocet | |
| • | (sometimes called Percs) | 14 |
| • | Prescription drugs not prescribed to you | 14 |
| _ | No | |
| П | Yes | |
| People | who experience discrimination may be at higher risk of negative health outcomes. Sha | ring your |
| | ences with discrimination in everyday life and in healthcare settings may help researche | |
| - | reduce negative health outcomes associated with discrimination. | |
| | - | |
| The next 3 statements describe how others may treat you. | | | | | | |
|---|---|--|--|--|--|--|
| In your day-to-day life, how often do any of these happen to you? | | | | | | |
| You are treated with less respect than other people are. | | | | | | |
| □ Never | | | | | | |
| ☐ Less than once a year | | | | | | |
| ☐ A few times a year | 15 | | | | | |
| ☐ A few times a month | | | | | | |
| ☐ At least once a week | | | | | | |
| ☐ Almost every day | | | | | | |
| People act as if they're better than you. | | | | | | |
| □ Never | | | | | | |
| ☐ Less than once a year | | | | | | |
| ☐ A few times a year | 16 | | | | | |
| ☐ A few times a month | 10 | | | | | |
| ☐ At least once a week | | | | | | |
| ☐ Almost every day | | | | | | |
| What do you think is the main reason for these experiences? (Select 1) | | | | | | |
| ☐ Your gender | | | | | | |
| ☐ Your sexual orientation | | | | | | |
| ☐ Your race | 17 | | | | | |
| ☐ Your religion | 17 | | | | | |
| ☐ Some aspect of your physical appearance | | | | | | |
| ☐ Your education or income level | | | | | | |
| ☐ Other: [Write in] | | | | | | |
| End Message: Thank you for completing this survey! | | | | | | |
| Persistence Assessment | | | | | | |
| Activity Title: Are You Still Taking PrEP? | | | | | | |
| Activity Description: In this short survey, we'll ask you some questions about your PrEI | journey | | | | | |
| and any challenges you may have encountered. | | | | | | |
| Activity: | | | | | | |
| 1. Are you still getting PrEP medicine by an injection from your healthcare provide | der? | | | | | |
| <ul><li>Yes, I am taking PrEP (branching logic to question 4)</li></ul> | | | | | | |
| ☐ No, I stopped taking PrEP (branching logic to question 2) | | | | | | |
| 2. If you stopped taking PrEP, which of the following best describes the reason(s | ) why? | | | | | |
| [Select up to 2] | , wily: | | | | | |
| | المملم الا | | | | | |
| ☐ I no longer feel I needed to take PrEP (branching logic to question 3 if se | iectea) | | | | | |
| It was too difficult to take to take PrEP as prescribed with my lifestyle | | | | | | |
| <ul> <li>I felt I was being judged by others for taking PrEP</li> </ul> | | | | | | |
| ☐ I experienced side effects from taking PrEP | | | | | | |

| | □ I take too many medications |
|---|---|
| | ☐ There were too many appointments as part of my PrEP care |
| | □ I tested positive for HIV |
| | □ Other: [Fill in the blank] |
| 3. Wh | ich of the following best describes why you no longer feel you need to take PrEP? |
| | □ I am no longer having sex |
| | □ I am in a monogamous relationship |
| | □ I am no longer using injectable drugs |
| | ☐ My partners and I are all regularly using condoms and getting tested for HIV |
| | □ Other: [Fill in the blank] |
| 4. If yo | ou are still taking PrEP, what challenges have you experienced? |
| | ☐ Have not experienced any challenges |
| | <ul> <li>Keeping up with clinical visits and laboratory testing</li> </ul> |
| | □ Concerns about side effects |
| | ☐ Finding transportation to my appointments |
| | <ul> <li>Stigma or discrimination from family, friends, or partner(s)</li> </ul> |
| | <ul> <li>Stigma or discrimination from healthcare professionals</li> </ul> |
| | □ Other: [Fill in the blank] |
| | a healthcare provider (for example, a doctor, nurse or pharmacist) or navigator |
| | r ask you what may make it difficult for you to take PrEP? (Month 1 & 11) — Yes |
| | □ No<br>□ Unsure |
| | □ Offsure |
| | <u>pe</u> : Patient Reported Outcomes – Set 1 |
| | le: Your Experiences With PrEP |
| | scription: This month we'll ask you to answer questions about your experience using |
| • | our thoughts about PrEP-related stigma. We'll also ask some questions about your using this mobile app to support you taking PrEP. The survey is 3 parts with a total |
| • | ions. It should take you 10-15 minutes to complete. |
| Activity: | nons. It should take you to is initiates to complete. |
| | us about your experience using PrEP |
| The followi | ng questions are related to the PrEP medicine you use to protect you from HIV |
| | nd your experience over the past 4 weeks. Please answer each question by selecting |
| | on each of the scales. |
| | satisfied are you with your <b>current medicine</b> for PrEP? |
| | Very satisfied |
| | Satisfied |

| | | Neither satisfied or dissatisfied |
|---|---|---|
| | | Dissatisfied |
| | | Very dissatisfied |
| 2. | Ho | w bothered are you by any side effects from the medicine you use for PrEP? |
| | | Very unbothered |
| | | Unbothered |
| | | Neither unbothered or bothered |
| | | Bothered |
| | | Very bothered |
| | | I have not experienced any side effects in the last 4 weeks |
| 3. | Ho | w satisfied are you with the <b>convenience</b> of PrEP recently? |
| | | Very satisfied |
| | | Satisfied |
| | | Neither satisfied or dissatisfied |
| | | Dissatisfied |
| | | Very dissatisfied |
| 4. | Ho | w satisfied are you with the <b>discreetness</b> of PrEP recently?<br>Very satisfied |
| | | Satisfied |
| | | Neither satisfied or dissatisfied |
| | | Dissatisfied |
| | | Very dissatisfied |
| 5. | Ho | w satisfied are you with your <b>understanding of using PrEP</b> to prevent HIV?<br>Very satisfied |
| | | Satisfied |
| | | Neither satisfied or dissatisfied |
| | | Dissatisfied |
| | | Very dissatisfied |
| 6. | Ho | w satisfied are you with the extent to which PrEP fits in with your lifestyle? |
| | | Very satisfied |
| | | Satisfied |
| | | Neither satisfied or dissatisfied |
| | | Dissatisfied |
| | | Very dissatisfied |
| 7. | Wo | ould you recommend this type of PrEP to someone else who wants to protect themselves from HIV? |

| | Ш | res, I would <b>definitely recommend</b> this type of Prep |
|----|----|------------------------------------------------------------------|
| | | Yes, I would <b>recommend</b> this type of PrEP |
| | | Not sure if I would recommend or not recommend this type of PrEP |
| | | No, I would <b>not recommend</b> this type of PrEP |
| | | No, I would <b>definitely not recommend</b> this type of PrEP |
| 8. | Ho | w satisfied would you be to continue your present form of PrEP? |
| | | Very satisfied |
| | | Satisfied |
| | | Neither satisfied or dissatisfied |
| | | Dissatisfied |
| | | Very dissatisfied |

# Part 2. What are your thoughts about PrEP-related stigma?

Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute. Please answer the following statements to the best of your ability.

# Indicate how much you agree with the following:

| | Completely agree | Agree | Neither agree<br>or disagree | Disagree | Completely disagree |
|---|---|---|---|---|---|
| I feel ashamed to go to the doctor for PrEP injections/shots. | () | () | () | () | () |
| People experience negative judgment because they take PrEP. | () | () | () | () | () |
| Someone using PrEP should keep their PrEP injection appointments hidden. | () | () | () | () | () |

| | Completely<br>agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| Someone taking PrEP would be seen by others as slutty. | () | () | () | () | () |

| People taking PrEP receive praise for being responsible. | () | () | () | () | () |
|---|---|---|---|---|---|
| My friends would be supportive of me taking PrEP. | () | () | () | () | () |

| | Completely<br>agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| Someone taking PrEP would be treated unfairly by their doctors. | () | () | () | () | () |
| People experience problems when they tell their sex partner(s) they are taking PrEP. | () | () | () | () | () |
| I feel proud to take PrEP. | () | () | () | () | () |

| | Completely<br>agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| People on PrEP are taking care of their health. | () | () | () | () | () |
| My family would be supportive of me taking PrEP. | () | () | () | () | () |

# Part 3. What is your experience using the TheraPay mobile app?

Please assess your experience using the TheraPay mobile app to support you in your journey using PrEP.

| | Completely agree | Agree | Neither<br>agree nor<br>disagree | Disagree | Completely disagree |
|---|---|---|---|---|---|
| 1. The TheraPay mobile app meets my approval. | 1 | 2 | 3 | 4 | 5 |
| 2. The TheraPay mobile app is appealing to me. | 1 | 2 | 3 | 4 | 5 |
| 3. I like the TheraPay mobile app. | 1 | 2 | 3 | 4 | 5 |
| 4. I welcome the TheraPay mobile app. | 1 | 2 | 3 | 4 | 5 |

**End Message:** Thank you for completing this survey! We will ask you these same questions again later to see how your responses have changed.

# Patient Reported Outcomes – Set 2

**Activity Title:** Your Experiences With PrEP

<u>Activity Description:</u> This month we'll ask you to answer questions about your experience using PrEP (pre-exposure prophylaxis). We'll also ask some questions about your experience using this mobile app to support you taking PrEP. The survey is two parts with a total of 16 questions. It should take you 8-12 minutes to complete.

Part 1. Tell us about your experience using PrEP

| Question | Question #<br>CAB LA Arm<br>[14] | Sub-concept |
|---|---|---|
| Over the past 4 weeks, how confident were you that PrEP prevented you from acquiring HIV? Very confident Quite confident Somewhat confident A little confident Not at all confident | 1 | Perceived efficacy |
| [CAB-LA arm] Over the past 4 weeks, did you experience any side effects, including injection site side effects (such as redness, bruising, or swelling) from the PrEP injection? □ No (branching logic to question 5) □ Yes (branching logic to show 3) | 2 | Acceptance of side effects |
| Over the past 4 weeks, how acceptable or unacceptable did you find the side effects from PrEP? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable Very unacceptable | 3<br>(branching<br>logic) | Acceptance of side effects |
| Over the past 4 weeks, did the side effects of the PrEP medication interfere with your physical activity (such as lifting things, walking, jogging), your leisure or free time activities (such as gardening, reading, dancing, visiting friends), or your daily activities (such as shopping, working, house work, yard work)? No, not at all Yes, a little Yes, somewhat Yes, quite a bit Yes, very much | 4 (branching<br>logic) | Acceptance of side<br>effects |
| [CAB LA arm] Over the past 4 weeks, did you experience any pain when getting your PrEP injection? | 5 | Acceptance of side effects |

| □ No (branching logic to question 7) | | |
|---|---|---|
| ☐ Yes (branching logic to question 6) [CAB LA arm] Over the past 4 weeks, how acceptable or | | |
| unacceptable did you find the <b>pain</b> you experienced when getting your PrEP injection? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable Very unacceptable | 6<br>(branching<br>logic) | Acceptance of side<br>effects |
| [CAB LA arm] Over the past 4 weeks, how acceptable or | | |
| unacceptable did you find the time it took to get the PrEP injection at your doctor's office? | | |
| <ul> <li>□ Very acceptable</li> <li>□ Acceptable</li> <li>□ Neither acceptable or unacceptable</li> <li>□ Unacceptable</li> <li>□ Very unacceptable</li> </ul> | 7 | Convenience |
| [CAB LA arm] Over the past 4 weeks, how acceptable or unacceptable did you find the number of times you had to get your PrEP injection? | | |
| <ul> <li>□ Very acceptable</li> <li>□ Acceptable</li> <li>□ Neither acceptable or unacceptable</li> <li>□ Unacceptable</li> <li>□ Very unacceptable</li> </ul> | 8 | Convenience |
| [CAB LA arm] Over the past 4 weeks, how easy or difficult was it to remember to go to your appointments for your PrEP injection? | | |
| <ul> <li>□ Very easy</li> <li>□ Easy</li> <li>□ Neither easy or difficult</li> <li>□ Difficult</li> <li>□ Very difficult</li> </ul> | 9 | Convenience |

| to fit in getting the PrEP injection into your daily life? Very easy Easy 10 Convenience Neither easy or difficult Difficult Very difficult Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? No, not at all Yes, octasionally 11 Convenience Yes, often Yes, often Yes, all the time Yes yer convenient Yes yer convenient Yes yer convenient Yes yer convenient Yes yer inconvenient Yes yer probably Yes yer babbly not Yes definitely Yes probably not Definitely not Probably not Definitely not Probably not Definitely not Yes, probably Yes, definitely Yes, definitely Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, definitely Yes, definitely Yes, definitely Yes, definitely Yes, probably Yes, definitely | [CAB LA arm] Over the past 4 weeks, how easy or difficult was it | | |
|---|---|---|---|
| Easy Neither easy or difficult Difficult Very difficult Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? No, not at all Yes, occasionally Yes, occasionally Yes, occasionally Yes, all the time Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Neither convenient or inconvenient Inconvenient Very inconvenient Very inconvenient Very inconvenient Very inconvenient Inconvenient Very inconvenient Very i | to fit in getting the PrEP injection into your daily life? | | |
| Neither easy or difficult Difficult Difficult Very difficult Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? No, not at all Yes, occasionally No, not at all Yes, octan Yes, other Yes, other Yes, all the time Yery convenient Yery convenient Yery convenient Yery inconvenient Yery inconvenient Yery inconvenient Yery inconvenient Yery inconvenient Yes definitely Yes probably not Definitely not Probably not Definitely not Definitely not Definitely not Definitely not Definitely not Yes, probably Yes, probably Yes, probably Yes, probably Yes, probably Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, deceptable Neither acceptable Neither acceptable or unacceptable Neither acceptable Neither acce | □ Very easy | | |
| Difficult □ Very difficult □ Very difficult Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? □ No, not at all □ Yes, occasionally □ Yes, octasionally □ Yes, often □ Yes, quite often □ Yes, all the time Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? □ Very convenient □ Convenient □ Neither convenient or inconvenient □ Inconvenient □ Very inconvenient □ Very inconvenient □ Yes definitely □ Yes probably □ I don't know □ Probably not □ Definitely not □ Probably not □ Definitely not □ Probably not □ I don't know □ Horobably not □ Probably not □ | □ Easy | 10 | Convenience |
| □ Very difficult Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? | ☐ Neither easy or difficult | | |
| Over the past 4 weeks, did you ever feel like you needed to hide your attendance to PrEP injection appointments so others would not see you? No, not at all Yes, occasionally Yes, often Yes, quite often Yes, all the time Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Neither convenient or inconvenient Inconvenient Very inconvenient Yes probably Yes definitely Yes probably Yes probably Definitely not Definitely not Definitely not Probably not Definitely not Defini | □ Difficult | | |
| your attendance to PrEP injection appointments so others would not see you? No, not at all Yes, occasionally Yes, outte often Yes, guite often Yes, all the time Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Neither convenient or inconvenient Inconvenient Very inconvenient Yes definitely Yes probably I don't know Probably not Definitely not Definitely not Definitely not Probably not Definitely not Definitely not Neither convenient or inconvenient I don't know Prespobably not Definitely not Neither acceptable Neither acceptable did you find the medicine? Very acceptable Neither acceptable | □ Very difficult | | |
| not see you? No, not at all Yes, occasionally Yes, often Yes, all the time Ves, all the time Ves, all the time Ves, all the time Ves, all the time Very convenient or inconvenient did you find taking the PrEP? Very convenient Convenient 12 | | | |
| No, not at all Yes, occasionally Yes, often Yes, quite often Yes, quite often Yes, all the time Yes, onvenient Yery convenient Yery convenient Yery convenient Yery inconvenient Yery inconvenient Yes probably Yes, and the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Yes probably Yes, probably Yes, probably Yes, probably Yes, definitely Yes, probably Yes, definitely Yes, def | | | |
| Yes, occasionally Yes, often Yes, quite often Yes, all the time Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Inconvenient Very inconvenient Very inconvenient Very inconvenient Icab La arm] In the future, would you choose to continue using the PrEP injection to protect yourself from HIV infection? Yes definitely Yes probably Idon't know Probably not Definitely not Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Icab La arm] In the future, would you choose to switch to using | | | |
| Yes, octain Yes, octain Yes, often Yes, quite often Yes, all the time Yes, all the past 4 weeks, how convenient or inconvenient 12 | | 11 | Convenience |
| Yes, quite often Yes, all the time Yes, all the time | | | |
| Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Neither convenient or inconvenient Inconvenient Very inconvenient Very inconvenient Idon't know Probably not Definitely not Definitely not Probably not Definitely not Vers, definitely Yes, probably Graph of Prep pill to protect yourself from HIV infection? Definitely not Probably not Vers, definitely Ves, definitely Ves, definitely Overall Acceptance Overall Acceptance Overall Acceptance Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable Acceptable Neither acceptable Neither acceptable Unacceptable Unacceptable Unacceptable Unacceptable Overall Acceptance | | | |
| Over the past 4 weeks, how convenient or inconvenient did you find taking the PrEP? Very convenient Convenient Neither convenient or inconvenient Inconvenient Very inconvenient Very inconvenient CAB LA arm] In the future, would you choose to continue using the PrEP injection to protect yourself from HIV infection? Yes definitely Probably I don't know Probably not Definitely not PreP pill to protect yourself from HIV infection? CAB LA arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Definitely not Probably not I don't know Yes, probably Yes, definitely Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable Acceptable Neither acceptable Neither acceptable Unacceptable Unacceptable Unacceptable | | | |
| find taking the PrEP? | | | |
| Convenient Neither convenient or inconvenient Inconvenient Very inconvenient CAB LA arm] In the future, would you choose to continue using the PrEP injection to protect yourself from HIV infection? Yes definitely Yes probably I don't know Probably not Definitely not CAB LA arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? I don't know Probably not Definitely not I don't know Yes, probably Yes, definitely Yes, definitely Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Neither acceptable or unacceptable Unacceptable Unacceptable Unacceptable Unacceptable | <u> </u> | | |
| Neither convenient or inconvenient 12 Convenience | □ Very convenient | | |
| Neither convenient or inconvenient Inconvenient Inconvenient Very inconvenient Very inconvenient | ☐ Convenient | 12 | Convenience |
| Very inconvenient | ☐ Neither convenient or inconvenient | 12 | Convenience |
| [CAB LA arm] In the future, would you choose to continue using the PrEP injection to protect yourself from HIV infection? Yes definitely | ☐ Inconvenient | | |
| the PrEP injection to protect yourself from HIV infection? Yes definitely Yes probably I don't know Probably not Definitely not [CAB LA arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Definitely not Probably not I don't know Yes, probably Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable Unacceptable Unacceptable Unacceptable Unacceptable | □ Very inconvenient | | |
| Yes probably | | | |
| Yes probably | ☐ Yes definitely | | |
| I don't know Probably not Definitely not | | 13 | Overall Acceptance |
| CAB LA arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Definitely not Probably not I don't know Yes, probably Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable Unacceptable Unacceptable | | - | |
| CAB LA arm] In the future, would you choose to switch to using the PrEP pill to protect yourself from HIV infection? Definitely not Probably not I don't know Yes, probably Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable Unacceptable Unacceptable | ☐ Probably not | | |
| the PrEP pill to protect yourself from HIV infection? Definitely not Probably not I don't know Yes, probably Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable Unacceptable Unacceptable | <u> </u> | | |
| □ Probably not □ I don't know □ Yes, probably □ Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? □ Very acceptable □ Acceptable □ Neither acceptable □ Unacceptable □ Unacceptable | | | |
| □ Probably not □ I don't know □ Yes, probably □ Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? □ Very acceptable □ Acceptable □ Neither acceptable □ Unacceptable □ Unacceptable | ☐ Definitely not | | |
| ☐ I don't know ☐ Yes, probably ☐ Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? ☐ Very acceptable ☐ Acceptable ☐ Neither acceptable ☐ Unacceptable ☐ Unacceptable | | 14 | Overall Acceptance |
| Yes, probably Yes, definitely Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable Unacceptable Unacceptable | <u> </u> | | |
| Thinking about all aspects of using PrEP over the past 4 weeks, how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable Unacceptable | | | |
| how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable | ☐ Yes, definitely | | |
| how acceptable or unacceptable did you find the medicine? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable | Thinking about all aspects of using DrED over the past 4 weeks | | |
| <ul> <li>□ Very acceptable</li> <li>□ Acceptable</li> <li>□ Neither acceptable or unacceptable</li> <li>□ Unacceptable</li> </ul> | | | |
| <ul> <li>□ Acceptable</li> <li>□ Neither acceptable or unacceptable</li> <li>□ Unacceptable</li> </ul> 15 Overall Acceptance □ Unacceptable | · | | |
| <ul><li>□ Neither acceptable or unacceptable</li><li>□ Unacceptable</li></ul> | | 15 | Overall Accentance |
| □ Unacceptable | · · | 13 | Overall Acceptance |
| | · | | |
| | ☐ Very unacceptable | | |

| did | erall, over the past 4 weeks, how acceptable or unacceptable you find taking all of your medicines, including PrEP and any per pills, tablets, or injections? | | |
|---|---|---|---|
| | Very acceptable | | |
| | Acceptable | 16 | Overall Acceptance |
| | Neither acceptable or unacceptable | | |
| | Unacceptable | | |
| | Very unacceptable | | |

Part 2. What is your experience using this mobile app?

Please assess how **appropriate** the use of a mobile app has been to support you in your journey using PrEP.

| | Completely agree | Agree | Neither<br>agree<br>nor<br>disagree | Disagree | Completely disagree |
|---|---|---|---|---|---|
| 1. Using a mobile app to support me using PrEP seems fitting. | 1 | 2 | 3 | 4 | 5 |
| 2. Using a mobile app to support me using PrEP seems suitable. | 1 | 2 | 3 | 4 | 5 |
| 3. Using a mobile app seems applicable. | 1 | 2 | 3 | 4 | 5 |
| 4. Using a mobile app to support me using PrEP seems like a good match. | 1 | 2 | 3 | 4 | 5 |

<u>End Message:</u> Thank you for completing this survey! We will ask you these same questions again later to see how your responses have changed.

**Health Literacy Evaluation - Month 2** 

Activity Description: Was the pop quiz on PrEP medicine helpful? What did you learn?

#### **Activity:**

1. How helpful was the pop quiz reviewing important facts about PrEP?



2. True/False: A person who takes PrEP will also need to use condoms to prevent other STIs.

#### □ True

 That's correct! PrEP only protects against HIV. Condoms will protect you against other sexually transmitted infections, such as syphilis, gonorrhea, or chlamydia.
 Condoms will also protect against unintended pregnancy.

#### □ False

 Not quite. PrEP only protects against HIV. Condoms will protect you against other sexually transmitted infections, such as syphilis, gonorrhea, or chlamydia.
 Condoms will also protect against unintended pregnancy.

#### **Health Literacy Evaluation – Month 4**

Activity Description: Was the video on protecting yourself helpful? What did you learn?

#### Activity:

1. How helpful was the video on sexual health, safer IV drug use, and protecting yourself?



# 2. True/False: All body parts used for sex should be tested for HIV & sexually transmitted infections (STIs).

#### □ True

That's correct! In many cases, this means you should have three body parts tested – (1) the throat; (2) the front (vagina, front hole, penis, urethra); and (3) the back (anus and rectum).

#### □ False

Not quite. All body parts used for sex should be tested for STIs. In many cases, this means you should have three body parts tested – (1) the throat; (2) the front (vagina, front hole, penis, urethra); and (3) the butt hole and rectum.

#### 3. True/False: All sexually transmitted infections (STIs) will cause symptoms.

#### a. True

Not quite. Many STIs do not cause any symptoms that you would notice. It is important to get regular testing.

#### b. False

That's correct! Many STIs do not cause any symptoms that you would notice. It is important to get regular testing.

#### **Health Literacy Evaluation – Month 6**

<u>Activity Description:</u> Was the video on "Building a Support System for HIV Prevention" helpful? What did you learn?

#### **Activity:**

1. How helpful was the video on building your support system?



- 2. True/False: West Virginia Health Right has services available if you are facing stressors or challenges.
- True That's right! There are many services available including telehealth appointments, health education classes, support for alcohol or drug addiction, LGBTQIA+ health, help from social workers, family planning services, dental and vision care, primary health care, behavioral or mental health care, pharmacy, and testing and screening for different health concerns. You can contact WVHR at 304-414-5930 for more
  - Not quite. There are many services available including telehealth appointments, health education classes, support for alcohol or drug addiction, LGBTQIA+ health, help from social workers, family planning services, dental and vision care, primary health care, behavioral or mental health care, pharmacy, and testing and screening for different health concerns. You can contact WVHR at 304-414-5930 for more information.
- 3. True/False: A support person could be a partner, family member, friend, peer navigator, or social worker.
  - ☐ **True**That's correct. Any one of these people could help support you. It's your choice and completely up to you who you want to bring on your support team.
    - Not quite. Any one of these people could help support you. It's your choice and completely up to you who you want to bring on your support team.

#### **Health Literacy Evaluation – Month 8**

☐ False

information.

□ False

<u>Activity Description:</u> Was the article on "Being an Active Participant in Your Own Care" helpful? What did you learn?

#### **Activity:**

#### 1. How helpful was the article on being an active participant in your own care?



- 2. Which of the following best describes shared decision-making?
  - When your doctor makes a decision about your healthcare that they feel is in your best interest

Not quite. Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

☐ When you and your doctor work together to make a decision about your healthcare that considers your values, goals and concerns

That's right! Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

☐ When your doctor works with another member of the care team (such as a nurse or social worker) to make a decision about your healthcare

Not quite. Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

- 3. True/False: Asking questions during your appointments is an important part of shared decision-making.
  - ☐ True

That's right! By asking your healthcare provider questions, you can get all of the information you need to make decisions about your health.

☐ False

Not quite. By asking your healthcare provider questions, you can get all of the information you need to make decisions about your health.

**Health Literacy Evaluation – Month 8** 

<u>Activity Description:</u> Was the video on "Overcoming Stigma and Becoming a Health Advocate" helpful? What did you learn?

#### **Activity:**

1. How helpful was the video on overcoming stigma and becoming a health advocate?



- 2. True/False: Stigma is when someone views a person or themselves in a negative way because of their unique identity, circumstances, and/or experiences.
  - True
     That's right! Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute.
    - □ False

      Not quite. Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute.
- 3. True/False: Sharing your experience with PrEP can help fight stigma surrounding it.
  - □ **True**That's right! Calling out biases and finding support within a community can help break the stigma cycle.
    - Not quite. Calling out biases and finding support within a community can help break the stigma cycle.

□ False

# Appendix C: Oral PrEP Arm Instruments

**<u>Activity Title</u>**: Baseline Information About You

Activity Description: Today we'll ask you to answer some questions about yourself. The survey

is 17 questions and should take about 10 minutes to complete.

# **Baseline Demographic Survey**

| Question | Question # |
|---|---|
| What year were you born? [Write in] | 1 |
| Which of the following best describes your racial/ethnic background? (Select all that | |
| apply) | |
| ☐ African American/Black | |
| ☐ Asian/Pacific Islander | 2 |
| ☐ Caucasian/White | 2 |
| ☐ Hispanic/Latinx | |
| □ Native American/Alaska Native | |
| ☐ A race or ethnicity not listed: [Write in] | |
| How do you describe your gender? (Select 1) | |
| ☐ Female | |
| □ Male | |
| ☐ Transgender woman | 3 |
| ☐ Transgender man | |
| □ Non-binary | |
| ☐ A gender not listed: [Write in] | |
| How do you describe your sexual orientation? (Select 1) | |
| ☐ Heterosexual/Straight | |
| ☐ Gay or Lesbian | |
| ☐ Bisexual | 4 |
| ☐ Queer or Sexually Fluid | |
| □ Pansexual | |
| ☐ A sexual orientation not listed: [Write in] | |
| What is the highest degree or school level you have completed? (Select 1) | |
| ☐ Primary school | |
| ☐ Some high school | |
| ☐ High school diploma or GED | |
| ☐ Some college | 5 |
| ☐ 2-year college degree | |
| ☐ 4-year college degree | |
| ☐ Graduate level degree | |
| ☐ An school level not listed: [Write in] | |
| What health coverage are you currently enrolled with? (Select up to 2) | |
| ☐ Medicaid | |
| ☐ Medicare | 6 |
| ☐ Affordable Care Act | 6 |
| ☐ Uninsured | |
| ☐ Private health insurance | |

| ☐ A health coverage not listed: [Write in] | |
|---|---|
| Why are using pre-exposure prophylaxis (PrEP) to prevent HIV? [Select all that apply] | |
| ☐ Reduce acquisition of HIV from sex | 7 |
| ☐ Reduce acquisition of HIV from IV drug use | |
| The next 5 questions ask about your food, housing, and transportation routines from th | e past 12 months. |
| If you have concerns and need support, please check in with your provider at your next | - |
| for immediate support. | |
| In the last 12 months, was there a time when you were not able to pay the mortgage or | |
| rent on time? | |
| □ No | 8 |
| □ Yes | |
| ☐ Not applicable | |
| In the last 12 months, was there a time when you did not have a steady place to sleep or | |
| slept in a shelter (including now)? | |
| □ No | 9 |
| □ Yes | |
| In the last 12 months, have you or the people you live with been unable to get utilities | |
| (heat, electricity) when it was really needed? | |
| □ No | 10 |
| □ Yes | |
| Within the past 12 months, the food you bought just didn't last and you didn't have | |
| money to get more. | |
| □ Never true | 11 |
| □ Sometimes true | |
| □ Often true | |
| Within the past 12 months, has lack of transportation kept you from medical | |
| appointments, getting your medicines, non-medical meetings or appointments, work, or | |
| from getting things that you need? | 12 |
| □ No | |
| □ Yes | |
| Do you feel physically and emotionally safe where you currently live? | |
| □ Yes | 13 |
| □ No | |
| During the past 30 days, have you used any of the following? | |
| An illegal drug (such as by snorting it or injecting it) | |
| Pain killer to get high (like OxyContin, sometimes called Oxy or OC) or Percocet | |
| (sometimes called Percs) | 14 |
| Prescription drugs not prescribed to you | |
| □ No | |
| □ Yes | |
| People who experience discrimination may be at higher risk of negative health outcomes. | l<br>Sharing vour |
| experiences with discrimination in everyday life and in healthcare settings may help resear | |
| reduce negative health outcomes associated with discrimination. | |
| The next 3 statements describe how others may treat you. | |

| | ay-to-day life, how often do any of these happen to you? | |
|---|---|---|
| You are tr | eated with less respect than other people are. | |
| | ever | |
| | ess than once a year | |
| □ A | few times a year | 15 |
| □ A | few times a month | 13 |
| □ A | t least once a week | |
| □ A | lmost every day | |
| People ac | t as if they're better than you. | |
| □ N | ever | |
| | ess than once a year | |
| □ A | few times a year | 16 |
| □ A | few times a month | 16 |
| □ A | t least once a week | |
| □ A | lmost every day | |
| What do | you think is the main reason for these experiences? (Select 1) | |
| | our gender | |
| | our sexual orientation | |
| | our race | |
| | our religion | 17 |
| | ome aspect of your physical appearance | |
| | our education or income level | |
| | ther: [Write in] | |
| | age: Thank you for completing this survey! | |
| Persisten | ce Assessment | |
| Activity Ti | tle: Are You Still Taking PrEP? | |
| | <u>escription:</u> In this short survey, we'll ask you some questions about your P | rEP iournev |
| | nallenges you may have encountered. | , |
| Activity: | idiiciiges you may nave encountered. | |
| | e you still taking PrEP medicine by mouth? | |
| | ☐ Yes, I am taking PrEP (branching logic to question 4) | |
| | □ No, I stopped taking PrEP (branching logic to questions 2) | |
| | 10, 1 stopped taking 1 Er (ordinating logic to questions 2) | |
| 2. Ov | er the past week, how many days did you miss taking PrEP? | |
| | 0 | |
| | 1 | |
| | 2 | |
| П | 3 | |
| | 4 | |
| Ц | 5 | |
| П | 6 | |

| | $\square$ 7 |
|---|---|
| 3. | If you stopped taking PrEP, which of the following best describes the reason(s) why? |
| | [Select up to 2] |
| | ☐ I no longer feel I needed to take PrEP (branching logic to question 3 if selected) |
| | ☐ It was too difficult to take PrEP with my schedule |
| | $\ \square$ I did not want people to know I was taking it or I felt I was being judged by |
| | others for taking PrEP |
| | ☐ I did not like the side effects |
| | ☐ I take too many medications |
| | ☐ There were too many appointments as part of my PrEP care |
| | ☐ I tested positive for HIV |
| | ☐ Other: [Fill in the blank] |
| 4. | Which of the following best describes why you no longer feel you need to take PrEP? |
| | ☐ I am no longer having sex |
| | ☐ I am in a monogamous relationship |
| | ☐ I am no longer using injectable drugs |
| | ☐ My partners and I are all regularly using condoms and getting tested for HIV |
| | ☐ Other: [Fill in the blank] |
| 5. | If you are still taking PrEP, what challenges have you experienced? [Select up to 2] |
| | ☐ Have not experienced any challenges |
| | ☐ Remembering to take PrEP every day |
| | ☐ Keeping up with clinical visits and laboratory testing |
| | ☐ Concerns about side effects |
| | ☐ Finding transportation to my appointments |
| | <ul> <li>Stigma or discrimination from family, friends, or partner(s)</li> </ul> |
| | ☐ Stigma or discrimination from healthcare professionals |
| | ☐ Other: [Fill in the blank] |
| 6. | Did a healthcare provider (for example, a doctor, nurse, or pharmacist) or navigator |
| | ever ask you what may make it difficult for you to take PrEP? |
| | □ Yes |
| | □ No |
| | □ Unsure |
| End M | essage: Thank you for completing this survey! |

Patient Reported Outcomes – Set 1

<u>Activity Title</u>: Your Experiences with PrEP

<u>Activity Description:</u> This month we'll ask you to answer questions about your experience using PrEP and your thoughts about PrEP-related stigma. We'll also ask some questions about your experience using this mobile app to support you taking PrEP. The survey is 3 parts with a total of 24 questions. It should take you 10-15 minutes to complete.

### **Activity:**

#### Part 1. Tell us about your experience using PrEP

The following questions are related to the PrEP medicine you use to protect you from HIV infection and your experience over the **past 4 weeks.** Please answer each question by selecting a number on each of the scales.

| 1. | Hov | v sat | isfied are you with your <b>current medicine</b> for PrEP? |
|---|---|---|---|
| | | | Very satisfied |
| | | | Satisfied |
| | | | Neither satisfied or dissatisfied |
| | | | Dissatisfied |
| | | | Very dissatisfied |
| 2. | Hov | v <b>bo</b> t | thered are you by any side effects from the medicine you use for PrEP? |
| | | Ver | y unbothered |
| | | Unb | oothered |
| | | Neit | ther unbothered or bothered |
| | | Botl | nered |
| | | Ver | y bothered |
| | | I ha | ve not experienced any side effects in the last 4 weeks |
| 3. | Hov | v sat | isfied are you with the <b>convenience</b> of PrEP recently? |
| | | Ver | y satisfied |
| | | Sati | sfied |
| | | Neit | ther satisfied or dissatisfied |
| | | Diss | atisfied |
| | | Ver | y dissatisfied |
| 4. | Hov | | isfied are you with the <b>discreetness</b> of PrEP recently?<br>y satisfied |
| | | Sati | sfied |
| | | Neit | ther satisfied or dissatisfied |
| | | Diss | atisfied |
| | | Ver | y dissatisfied |
| 5. | Hov | v sat | isfied are you with your <b>understanding of using PrEP</b> to prevent HIV?<br>Very satisfied |
| | | | Satisfied |

| | | | Neither satisfied or dissatisfied |
|---|---|---|---|
| | | | Dissatisfied |
| | | | Very dissatisfied |
| 6. | Hov | w sat | isfied are you with the extent to which PrEP fits in with your lifestyle? |
| | | | Very satisfied |
| | | | Satisfied |
| | | | Neither satisfied or dissatisfied |
| | | | Dissatisfied |
| | | | Very dissatisfied |
| 7. | Wo | Yes,<br>Yes,<br>Not | ou recommend this type of PrEP to someone else who wants to protect themselves from HIV? I would definitely recommend this type of PrEP I would recommend this type of PrEP sure if I would recommend or not recommend this type of PrEP I would not recommend this type of PrEP I would definitely not recommend this type of PrEP |
| 8. | Hov | w sat | isfied would you be to continue your present form of PrEP? |
| | | Ver | y satisfied |
| | | Sati | sfied |
| | | Nei | ther satisfied or dissatisfied |
| | | Diss | atisfied |
| | | Ver | y dissatisfied |

# Part 2. What are your thoughts about PrEP-related stigma?

Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute. Please answer the following statements to the best of your ability.

# Indicate how much you agree with the following:

| | Completely agree | Agree | Neither Agree<br>or Disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| I feel ashamed to take PrEP pills in front of others. | () | () | () | () | () |
| People experience negative judgment because they take PrEP. | () | () | () | () | () |

| Someone taking PrEP should keep their pills hidden. | () | () | () | () | () |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| | Completely<br>agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| Someone taking PrEP would be seen by others as slutty. | () | () | () | () | () |
| People taking PrEP receive praise for being responsible. | () | () | () | () | () |
| My friends would be supportive of me taking PrEP. | () | () | () | () | () |

| | Completely<br>agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| Someone taking PrEP would be treated unfairly by their doctors. | () | () | () | () | () |
| People experience problems when they tell their sex partner(s) they are taking PrEP. | () | () | () | () | () |
| I feel proud to take PrEP. | () | () | () | () | () |

| | Completely agree | Agree | Neither<br>agree or<br>disagree | Disagree | Completely<br>disagree |
|---|---|---|---|---|---|
| People on PrEP are taking care of their health. | () | () | () | () | () |
| My family would be supportive of me taking PrEP. | () | () | () | () | () |

# Part 3. What is your experience using the TheraPay mobile app?

Please assess your experience using the TheraPay mobile app to support you in your journey using PrEP.

| | Completely agree | Agree | Neither<br>agree nor<br>disagree | Disagree | Completely disagree |
|---|---|---|---|---|---|
| 1. The TheraPay mobile app meets my approval. | 1 | 2 | 3 | 4 | 5 |
| 2. The TheraPay mobile app is appealing to me. | 1 | 2 | 3 | 4 | 5 |
| 3. I like the TheraPay mobile app. | 1 | 2 | 3 | 4 | 5 |
| 4. I welcome the TheraPay mobile app. | 1 | 2 | 3 | 4 | 5 |

### Patient Reported Outcomes – Set 2

**Activity Title:** Your Experiences With PrEP

<u>Activity Description:</u> This month we'll ask you to answer questions about your experience using PrEP (pre-exposure prophylaxis). We'll also ask some questions about your experience using this mobile app to support you taking PrEP. The survey is two parts with a total of 16 questions. It should take you 8-12 minutes to complete.

Part 1. Tell us about your experience using PrEP

| Question | Question #<br>Oral PrEP Arm<br>[13] | Sub-concept |
|---|---|---|
| Over the past 4 weeks, how confident were you that PrEP prevented you from acquiring HIV? Very confident Quite confident Somewhat confident A little confident Not at all confident | 1 | Perceived efficacy |
| [Oral PrEP arm] Over the past 4 weeks, did you experience any side effects from the PrEP pill? No (branching logic to question 5) Yes (branching logic to show 3) | 2 | Acceptance of side effects |
| Over the past 4 weeks, how acceptable or unacceptable did you find the side effects from PrEP? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable Very unacceptable | 3<br>(branching<br>logic) | Acceptance of side effects |
| Over the past 4 weeks, did the side effects of the PrEP medication interfere with your physical activity (such as lifting things, walking, jogging), your leisure or free time activities (such as gardening, reading, dancing, visiting friends), or your daily activities (such as shopping, working, house work, yard work)? □ No, not at all | 4<br>(branching<br>logic) | Acceptance of side effects |

| | T | T |
|---|---|---|
| □ Yes, a little | | |
| ☐ Yes, somewhat | | |
| ☐ Yes, quite a bit | | |
| ☐ Yes, very much | | |
| [Oral PrEP arm] Over the past 4 weeks, did you ever feel like you | | |
| needed to hide your PrEP pills so others would not see them? | | |
| ☐ No, not at all | | |
| ☐ Yes, occasionally | 5 | N/A |
| ☐ Yes, often | | • |
| ☐ Yes, quite often | | |
| ☐ Yes, all the time | | |
| [Oral PrEP arm] Over the past 4 weeks, how acceptable or unacceptable did you find the time it took to take your PrEP pill every day? Uery acceptable | 6 | Convenience |
| □ Acceptable | | |
| □ Neither acceptable or unacceptable | | |
| □ Unacceptable | | |
| □ Very unacceptable | | |
| unacceptable did you find the number of times you had to take your PrEP pill? Very acceptable Acceptable Neither acceptable or unacceptable Unacceptable Very unacceptable Oral PrEP arm] Over the past 4 weeks, how easy or difficult was it | 7 | Convenience |
| to remember to take your PrEP pills? | | |
| <ul> <li>□ Very easy</li> <li>□ Easy</li> <li>□ Neither easy or difficult</li> <li>□ Difficult</li> <li>□ Very difficult</li> </ul> | 8 | Convenience |
| [Oral PrEP arm] Over the past 4 weeks, how easy or difficult was it to fit in taking the PrEP pill into your daily life? | | |
| □ Very easy | | |
| □ Easy | 9 | Convenience |
| Neither easy or difficult | | |
| □ Difficult | | |
| □ Very difficult | | |
| Over the past 4 weeks, how <b>convenient or inconvenient</b> did you find | | |
| taking the PrEP? | 10 | Convenience |
| □ Very convenient | | 1 |

| | T | 1 |
|---|---|---|
| □ Neither convenient or inconvenient | | |
| □ Very inconvenient | | |
| [Oral PrEP arm] In the future, would you choose to continue using | | |
| the PrEP pill to protect yourself from HIV infection? | | |
| ☐ Yes, definitely | | |
| ☐ Yes, probably | 11 | Overall Acceptance |
| ☐ I don't know | | overall receptance |
| □ Probably not | | |
| ☐ Definitely not | | |
| [Oral PrEP arm] In the future, would you choose to switch to using | | |
| the PrEP injection to protect yourself from HIV infection? | | |
| ☐ Definitely not | | |
| ☐ Probably not | 12 | Overall Acceptance |
| ☐ I don't know | | |
| ☐ Yes, probably | | |
| ☐ Yes, definitely | | |
| Thinking about <b>all aspects of using PrEP</b> over the past 4 weeks, how | | |
| acceptable or unacceptable did you find the medicine? | | |
| ☐ Very acceptable | | |
| □ Acceptable | 13 | Overall Acceptance |
| □ Neither acceptable or unacceptable | | |
| □ Unacceptable | | |
| □ Very unacceptable | | |
| Overall, over the past 4 weeks, how acceptable or unacceptable did | | |
| you find taking all of your medicines, including PrEP and any other | | |
| pills, tablets, or injections? | | |
| □ Very acceptable | 14 | Overall Acceptance |
| □ Acceptable | | o veran / teceptance |
| □ Neither acceptable or unacceptable | | |
| □ Unacceptable | | |
| ☐ Very unacceptable | | |

# Part 2. What is your experience using this mobile app?

Please assess how **appropriate** the use of a mobile app has been to support you in your journey using PrEP.

| | Completely agree | Agree | Neither<br>agree<br>nor<br>disagree | Disagree | Completely disagree |
|---|---|---|---|---|---|
| 1. Using a mobile app to support me using PrEP seems fitting. | 1 | 2 | 3 | 4 | 5 |

| 2. Using a mobile app to support me using PrEP seems suitable. | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| 3. Using a mobile app seems applicable. | 1 | 2 | 3 | 4 | 5 |
| 4. Using a mobile app to support me using PrEP seems like a good match. | 1 | 2 | 3 | 4 | 5 |

**End Message:** Thank you for completing this survey! We will ask you these same questions again later to see how your responses have changed.

#### **Health Literacy Evaluation - Month 2**

Activity Description: Was the pop quiz on PrEP medicine helpful? What did you learn?

#### **Activity:**

1. How helpful was the pop quiz reviewing important facts about PrEP?



- 2. True/False: A person who takes PrEP will also need to use condoms to prevent other STIs.
  - □ True
    - That's correct! PrEP only protects against HIV. Condoms will protect you against other sexually transmitted infections, such as syphilis, gonorrhea, or chlamydia.
       Condoms will also protect against unintended pregnancy.
  - □ False
    - Not quite. PrEP only protects against HIV. Condoms will protect you against other sexually transmitted infections, such as syphilis, gonorrhea, or chlamydia.
       Condoms will also protect against unintended pregnancy.

#### **Health Literacy Evaluation – Month 4**

Activity Description: Was the video on protecting yourself helpful? What did you learn?

#### **Activity:**

1. How helpful was the video on sexual health, safer IV drug use, and protecting yourself?



- 2. True/False: All body parts used for sex should be tested for HIV & sexually transmitted infections (STIs).
  - □ True

That's correct! In many cases, this means you should have three body parts tested - (1) the throat; (2) the front (vagina, front hole, penis, urethra); and (3) the back (anus and rectum).

□ False

Not quite. All body parts used for sex should be tested for STIs. In many cases, this means you should have three body parts tested – (1) the throat; (2) the front (vagina, front hole, penis, urethra); and (3) the butt hole and rectum.

- 3. True/False: All sexually transmitted infections (STIs) will cause symptoms.
  - a. True

Not quite. Many STIs do not cause any symptoms that you would notice. It is important to get regular testing.

b. False

That's correct! Many STIs do not cause any symptoms that you would notice. It is important to get regular testing.

#### **Health Literacy Evaluation – Month 6**

<u>Activity Description:</u> Was the video on "Building a Support System for HIV Prevention" helpful? What did you learn?

#### **Activity:**

1. How helpful was the video on building your support system?



- 2. True/False: West Virginia Health Right has services available if you are facing stressors or challenges.
  - □ True

That's right! There are many services available including telehealth appointments, health education classes, support for alcohol or drug addiction, LGBTQIA+ health, help from social workers, family planning services, dental and vision care, primary health care, behavioral or mental health care, pharmacy, and testing and screening for different health concerns. You can contact WVHR at 304-414-5930 for more information.

#### □ False

Not quite. There are many services available including telehealth appointments, health education classes, support for alcohol or drug addiction, LGBTQIA+ health, help from social workers, family planning services, dental and vision care, primary health care, behavioral or mental health care, pharmacy, and testing and screening for different health concerns. You can contact WVHR at 304-414-5930 for more information.

3. True/False: A support person could be a partner, family member, friend, peer navigator, or social worker.

#### □ True

That's correct. Any one of these people could help support you. It's your choice and completely up to you who you want to bring on your support team.

#### ☐ False

Not quite. Any one of these people could help support you. It's your choice and completely up to you who you want to bring on your support team.

#### **Health Literacy Evaluation – Month 8**

<u>Activity Description:</u> Was the article on "Being an Active Participant in Your Own Care" helpful? What did you learn?

#### **Activity:**

How helpful was the article on being an active participant in your own care?



- 2. Which of the following best describes shared decision-making?
  - ☐ When your doctor makes a decision about your healthcare that they feel is in your best interest

Not quite. Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

☐ When you and your doctor work together to make a decision about your healthcare that considers your values, goals and concerns

That's right! Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

☐ When your doctor works with another member of the care team (such as a nurse or social worker) to make a decision about your healthcare

Not quite. Shared decision-making is a process where you and your healthcare providers work together to make decisions that reflect what's most important to you while making sure your medications are safe and effective.

3. True/False: Asking questions during your appointments is an important part of shared decision-making.

#### □ True

That's right! By asking your healthcare provider questions, you can get all of the information you need to make decisions about your health.

#### ☐ False

Not quite. By asking your healthcare provider questions, you can get all of the information you need to make decisions about your health.

#### **Health Literacy Evaluation – Month 8**

<u>Activity Description:</u> Was the video on "Overcoming Stigma and Becoming a Health Advocate" helpful? What did you learn?

#### **Activity:**

1. How helpful was the video on overcoming stigma and becoming a health advocate?



2. True/False: Stigma is when someone views a person or themselves in a negative way because of their unique identity, circumstances, and/or experiences.

#### □ True

That's right! Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute.

| | | | False Not quite. Stigma is a negative and unfair belief about someone because of a particular characteristic or attribute. |
|---|---|---|---|
| | 3. T | rue/F | alse: Sharing your experience with PrEP can help fight stigma surrounding it. |
| | | | <b>True</b> That's right! Calling out biases and finding support within a community can help break the stigma cycle. |
| | | | <b>False</b> Not quite. Calling out biases and finding support within a community can help break the stigma cycle. |
| | | | Appendix D: Clinician Instruments |
| PRO | OVIDE | R SUF | RVEY (Note: baseline survey) |
| | - | | agreeing to be part of this quality improvement project to improve care for those ing PrEP. Your responses will remain confidential and anonymous. |
| Par | t 1. In | forma | ation About You and Your Patients |
| 1. | What | t year | were you born? [Write in] |
| 2. | How | | u describe your gender (response optional)? [Select 1] male |
| | | Ma | ale |
| | | Tra | ansgender woman |
| | | Tra | ansgender man |
| | | . No | on-binary |
| | | Pro | efer not to answer |
| | | Αį | gender not listed: [Write in] |
| 3. | | h of t<br>apply) | he following best describes your racial/ethnic background (response optional)? (Select all |
| | | Af | rican American/Black |
| | | As | ian/Pacific Islander |
| | | Ca | ucasian/White |

| | | Hispanic/Latinx |
|---|---|---|
| | | Native American/Alaska Native |
| | | A race or ethnicity not listed: [Write in] |
| 4. | What is | s your role within the interprofessional team? [Select 1] |
| | | Physician |
| | | Physician assistant |
| | | Nurse practitioner |
| | | Nurse |
| | | Medical assistant |
| | | Pharmacist |
| | | Case manager |
| | | Social worker |
| | | Clinic administrative staff |
| | | A role on the interprofessional team not listed: [Write in] |
| 5. | What is | s your role in the clinic for providing long-acting cabotegravir to your patients? (Select all tha |
| | ,, | □ Prescribing |
| | | ☐ Medication procurement and/or dispensing |
| | | □ Administering injections |
| | | □ Patient scheduling |
| | | ☐ Coordinating clinic flow (i.e., room availability, nurse scheduling, availability of injection |
| | | during appointment, etc) |
| | | ☐ Providing wraparound services (i.e., transportation, housing support, mental health |
| | | resources, etc.) |
| | | ☐ Patient counseling |
| | | ☐ A role not listed: [write in] |
| | | eptability, Appropriateness, and Feasibility of Implementing Long-Acting Cabotegravir |
| mi | ections | |

# Acceptability of Intervention Measure (AIM)

| | Completely disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| 1. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>meets my approval. | 0 | 0 | 0 | 0 | 0 |

| 2. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>is appealing to me. | 0 | 0 | 0 | 0 | 0 |
|---|---|---|---|---|---|
| 3. I like our clinic process for providing longacting cabotegravir injections to our clients. | 0 | 0 | 0 | 0 | 0 |
| 4. I welcome our clinic process for providing long-acting cabotegravir injections to our clients. | 0 | 0 | 0 | 0 | 0 |

# Intervention Appropriateness Measure (IAM)

| | Completely<br>disagree | Disagree | Neither<br>agree<br>nor<br>disagree | Agree | Completely<br>agree |
|---|---|---|---|---|---|
| 1. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems fitting. | 0 | 0 | 0 | 0 | 0 |
| 2. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems suitable. | 0 | 0 | 0 | 0 | 0 |
| 3. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems applicable. | 0 | 0 | 0 | 0 | 0 |
| 4. Our clinic process for providing longacting cabotegravir injections to our clients seems like a good match. | 0 | 0 | 0 | 0 | 0 |

# Feasibility of Intervention Measure (FIM)

| | Completely<br>disagree | Disagree | Neither<br>agree<br>nor<br>disagree | Agree | Completely agree |
|---|---|---|---|---|---|
| 1. Long-term use of cabotegravir injections in our clinic seem implementable. | 0 | 0 | 0 | 0 | 0 |
| 2. Long-term use of cabotegravir injections in our clinic seem possible. | 0 | 0 | 0 | 0 | 0 |

| 3. Long-term use of cabotegravir injections in our clinic seem doable. | 0 | 0 | 0 | 0 | 0 |
|---|---|---|---|---|---|
| 4. Long-term use of cabotegravir injections in our clinic seem easy to continue. | 0 | 0 | 0 | 0 | 0 |

# Part 3. Barriers and Facilitators for Implementation of Long-Acting Cabotegravir for PrEP

| 1. | Ple | ase rate your confidence in <b>initiating</b> and <b>monitoring</b> long-acting cabotegravir for PrEP. |
|---|---|---|
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| 2. | Ple | ase rate your confidence in administering long-acting cabotegravir for PrEP. |
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| 3. | Ple | ase rate your confidence in <b>counseling</b> patients in HIV prevention, addressing barriers to |
| | usi | ng PrEP, and supporting persistence. |
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| ease | indi | cate how much you agree with the following: |

# Ple

| | Strongly<br>agree | Agree | Neutral | Disagree | Strongly<br>disagree |
|---|---|---|---|---|---|
| 4. People experience negative judgment because they take PrEP. | () | () | () | () | () |
| 5. Someone taking PrEP would be seen by others as slutty. | () | () | () | () | () |

()

()

| 6. People taking PrEP receive praise for being responsible. | () | () | () | () | |
|---|---|---|---|---|---|
| 7. Someone taking PrEP would be treated unfairly by their doctors. | () | () | () | () | |
| 8. What barriers do you forest [Select up to 2] Patient's ability to keep Patient's transportation Flagging/Clinic awarene Staffing resourcing for a Rescheduling missed in Patients acquiring HIV a Management of patient Patient injection/soren. 9. Which structural changes o implementation in your clir Increased coordination Purchasing new refrige Finding room space or Adjusting or extending Use of different staff fo Making transportation Expanding hours for inj Accommodating patien same-day appointment Other: [write in] 10. How helpful do you think you persistence with PrEP? Very helpful Somewhat helpful Somewhat helpful Neither helpful or use Somewhat unhelpful Very unhelpful | bimonthly apport of for bimonthly a less of missed visions clinic flow jections due to missed do ts with other ne- less or resources may lic? [Select up to with other deparators working around staff working ho or injections arrangements for ection visits (i.e. ts needing to re s) our clients will fi | pointments appointments its pose/visit eds help facilitate pose/visit eds help facilitate pose/visit eds help facilitate pose/visit eds help facilitate pose/visit eds help facilitate pose/visit eds | long-acting cab<br>harmacy)<br>ty<br>cipants<br>ing or during lui<br>ion visits (i.e. us | otegravir<br>nch breaks)<br>sing walk-in visit | ts, |

11. Do you have a preference for prescribing long-acting cabotegravir or daily oral PrEP?

| | □ Pre | fer long-acting cabotegravir |
|---|---|---|
| | □ Pre | fer oral daily PrEP |
| | □ No | preference |
| | | ely is it that your clinic will continue to offer cabotegravir following the completion of |
| | this stu | • |
| | | ry likely<br>newhat likely |
| | | utral |
| | | newhat unlikely |
| | | y unlikely |
| em | • | aking the time to complete this survey. Please provide your work email address. Your e tied to your survey responses and will only be used for the purposes of this quality nitiative. |
| ТН | | ork email address: [Write in] R COMPLETING THIS SURVEY. |
| PR | OVIDER SUR | VEY (Note: 6 months, 12 months and end of study) |
| | • | greeing to be part of this quality improvement project to improve care for those ng PrEP. Your responses will remain confidential and anonymous. |
| | rt 1. Informa | tion About You and Your Patients |
| Pa | | |
| <b>Pa</b><br>6. | What year | tion About You and Your Patients |
| <b>Pa</b><br>6. | What year | were you born? [Write in] u describe your gender? [Select 1] nale |
| <b>Pa</b><br>6. | What year How do yo Fei | were you born? [Write in] u describe your gender? [Select 1] nale |
| <b>Pa</b><br>6. | What year How do yo Fer Ma | were you born? [Write in] u describe your gender? [Select 1] nale |
| <b>Pa</b><br>6. | What year How do yo Fer Ma Tra | were you born? [Write in] u describe your gender? [Select 1] nale le nsgender woman |
| <b>Pa</b><br>6. | What year How do yo Fee Ma Tra No | were you born? [Write in] describe your gender? [Select 1] nale le nsgender woman nsgender man |
| <b>Pa</b><br>6. | What year How do yo Fer Ma Tra No | tion About You and Your Patients were you born? [Write in] u describe your gender? [Select 1] nale le nsgender woman nsgender man n-binary |
| <b>Pa</b> 6. 7. | What year How do yo Fer Ma Tra Tra No | were you born? [Write in] describe your gender? [Select 1] nale le nsgender woman n-binary fer not to answer |
| <b>Pa</b><br>6. | What year How do yo Fee Ma Tra No Pre A g | were you born? [Write in] describe your gender? [Select 1] nale le nsgender woman nsgender man n-binary fer not to answer ender not listed: [Write in] |
| <b>Pa</b> 6. 7. | What year How do yo Fer Ma Tra No Pre Ag Which of the | were you born? [Write in] u describe your gender? [Select 1] nale le nsgender woman nsgender man n-binary fer not to answer ender not listed: [Write in] ne following best describes your racial/ethnic background? (Select all that apply) |

| | | Hispanic/Latinx |
|---|---|---|
| | | Native American/Alaska Native |
| | | A race or ethnicity not listed: [Write in] |
| 9. | What is | s your role within the interprofessional team? [Select 1] |
| | | Physician |
| | | Physician assistant |
| | | Nurse practitioner |
| | | Nurse |
| | | Medical assistant |
| | | Pharmacist |
| | | Case manager |
| | | Social worker |
| | | Clinic administrative staff |
| | | A role on the interprofessional team not listed: [Write in] |
| 10. | . What is | s your role in the clinic for providing long-acting cabotegravir to your patients? (Select all that |
| | apply) | |
| | | □ Prescribing |
| | | ☐ Medication procurement and/or dispensing |
| | | □ Administering injections |
| | | □ Patient scheduling |
| | | ☐ Coordinating clinic flow (i.e., room availability, nurse scheduling, availability of injection |
| | | during appointment, etc) |
| | | ☐ Providing wraparound services (i.e., transportation, housing support, mental health |
| | | resources, etc.) |
| | | □ Patient counseling |
| | | ☐ A role not listed: [write in] |
| Paı | rt 2. Acc | eptability, Appropriateness, and Feasibility of Implementing Long-Acting Cabotegravir |

Injections

#### Acceptability of Intervention Measure (AIM) Neither Completely Completely Disagree agree nor Agree disagree agree disagree 1. Our clinic process for providing long-0 0 0 0 0 acting cabotegravir injections to our clients meets my approval.

| 2. Our clinic process for providing longacting cabotegravir injections to our clients is appealing to me. | 0 | 0 | 0 | 0 | 0 |
|---|---|---|---|---|---|
| 3. I like our clinic process for providing longacting cabotegravir injections to our clients. | 0 | 0 | 0 | 0 | 0 |
| 4. I welcome our clinic process for providing long-acting cabotegravir injections to our clients. | 0 | 0 | 0 | 0 | 0 |

# **Intervention Appropriateness Measure (IAM)**

| | on Appropriat | | W. C (13 1111) | | |
|---|---|---|---|---|---|
| | Completely<br>disagree | Disagree | Neither<br>agree<br>nor<br>disagree | Agree | Completely agree |
| 1. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems fitting. | 0 | 0 | 0 | 0 | 0 |
| 2. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems suitable. | 0 | 0 | 0 | 0 | 0 |
| 3. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems applicable. | 0 | 0 | 0 | 0 | 0 |
| 4. Our clinic process for providing long-<br>acting cabotegravir injections to our clients<br>seems like a good match. | 0 | 0 | 0 | 0 | 0 |

#### **Feasibility of Intervention Measure (FIM)**

| | cy or micerven | | - (, | | |
|---|---|---|---|---|---|
| | Completely<br>disagree | Disagree | Neither<br>agree<br>nor<br>disagree | Agree | Completely agree |
| 1. Long-term use of cabotegravir injections in our clinic seem implementable. | 0 | 0 | 0 | 0 | 0 |
| 2. Long-term use of cabotegravir injections in our clinic seem possible. | 0 | 0 | 0 | 0 | 0 |
| 3. Long-term use of cabotegravir injections in our clinic seem doable. | 0 | 0 | 0 | 0 | 0 |
| 4. Long-term use of cabotegravir injections in our clinic seem easy to continue. | 0 | 0 | 0 | 0 | 0 |

# Part 3. Barriers and Facilitators for Implementation of Long-Acting Cabotegravir for PrEP

| 13. | Please | rate your confidence in initiating and monitoring long-acting cabotegravir for PrEP. |
|---|---|---|
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| 14. | Please | rate your confidence in administering long-acting cabotegravir for PrEP. |
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| 15. | Please | rate your confidence in <b>counseling</b> patients in HIV prevention, addressing barriers to using |
| | PrEP, a | nd supporting persistence. |
| | | Very high |
| | | High |
| | | Moderate |
| | | Low |
| | | Very low |
| | | Not applicable |
| 16. | Please | rate the impact of providing long-acting cabotegravir injections for PrEP on your workload in |
| | clinic. | |
| | | Large increase in workload |
| | | Moderate increase in workload |
| | | No change in workload |
| | | Moderate decrease in workload |
| | | Large decrease in workload |
| 17. | | parriers have you observed with the implementation of long-acting cabotegravir for PrEP? |
| | [Select | up to 2] |
| | | Patient's ability to keep bimonthly appointments |
| | | Patient's transportation for bimonthly appointments |
| | | Flagging/Clinic awareness of missed visits |
| | | Staffing resourcing for clinic flow |
| | | Rescheduling missed injections |
| | | Patients acquiring HIV due to missed dose/visit |
|---|---|---|
| | | Management of patients with other needs |
| | | Patient injection/soreness |
| 18. | Which | structural changes or resources have been most helpful in facilitating long-acting |
| | cabote | gravir implementation in your clinic? [Select up to 2] |
| | | Increased coordination with other departments (i.e., pharmacy) |
| | | Purchasing new refrigerators |
| | | Finding room space or working around room availability |
| | | Adjusting or extending staff working hours |
| | | Use of different staff for injections |
| | | Making transportation arrangements for patient participants |
| | | Expanding hours for injection visits (i.e., visits in morning or during lunch breaks) |
| | | Accommodating patients needing to reschedule injection visits (i.e. using walk-in visits, |
| | | same-day appointments) |
| | | Other: [write in] |
| 19. | How co | ould the process for use of long-acting cabotegravir injections for PrEP be improved? [Select |
| | up to 2 | ] |
| | □ Inc | reased clinic staff |
| | □ Red | distribution of clinic duties to allow dedicated healthcare providers more time to support |
| | lon | g-acting cabotegravir processes |
| | □ Re | gular evaluation of LA-CAB processes for efficacy and potential problems |
| | □ Ad | ditional staff education/training |
| | □ Im <sub>l</sub> | prove documentation/EMR |
| | □ Im <sub>l</sub> | prove communication and care coordination within the clinical team |
| | □ Im <sub>l</sub> | prove communication with clients using PrEP (i.e. reminders of upcoming appointments, |
| | res | cheduling of missed appointments) |
| | □ Otl | ner: [fill in blank] |
| 20. | For par | ticipants who stopped taking long-acting injectable PrEP, which of the following best |
| | describ | es the most common reason(s) why? [Select up to 2] |
| | | ☐ They no longer have an indication or need for PrEP |
| | | ☐ They found it too difficult to take PrEP as prescribed with their lifestyle |
| | | ☐ They felt stigmatized by others for taking PrEP |
| | | ☐ They experienced side effects from taking PrEP |
| | | ☐ They take too many medications |
| | | ☐ They felt there were too many appointments as part of PrEP care |
| | | ☐ They tested positive for HIV |

| 21. | How how with Pr | | I do you think your clients find the TheraPay mobile health app in supporting persistence |
|---|---|---|---|
| | | | Very helpful |
| | | | Somewhat helpful |
| | | | Neither helpful or unhelpful |
| | | П | Somewhat unhelpful |
| | | | Very unhelpful |
| 22. | Do you | ı hav | e a preference for prescribing long-acting cabotegravir or daily oral PrEP? |
| | | Pre | fer long-acting cabotegravir |
| | | Pre | fer oral daily PrEP |
| | | No | preference |
| 23. | How lil | kely i | s it that your clinic will continue to offer cabotegravir following the completion of this |
| | study? | | |
| | | Ver | y likely |
| | | Son | newhat likely |
| | | Net | utral |
| | | Son | newhat unlikely |
| | | Ver | y unlikely |
| Tha | nk you | for to | aking the time to complete this survey. Please provide your work email address. Your |
| | | | e tied to your survey responses and will only be used for the purposes of this quality |
| imp | roveme | ent ir | nitiative. |
| | | W | ork email address: [Write in] |
| T11/ | NII VO | | D COMPLETING THIS SUDVEY |

## Appendix E: Incentive Mapping

## **Incentive Mapping for CAB-LA Arm**

| Time Frame | Activity | Incentive |
|------------|-----------------------------|-----------|
| Month 0 | Baseline Demographic Survey | \$20 |
| Month 1 | Persistence assessment | \$5 |
| | PRO Survey #1 | \$10 |
| Month 2 | Health Literacy Survey | \$10 |
| Month 3 | PRO Survey #2 | \$10 |
| | Persistence assessment | \$10 |
| Month 4 | Health Literacy Survey | \$10 |
| Month 5 | Persistence assessment | \$15 |
| | PRO Survey #1 | \$15 |
| Month 6 | Health Literacy Survey | \$10 |
| Month 7 | Persistence assessment | \$15 |
| Month 8 | Health Literacy Survey | \$10 |
| Month 9 | Persistence assessment | \$15 |
| | PRO Survey #2 | \$20 |
| Month 10 | Health Literacy Survey | \$10 |
| Month 11 | Persistence assessment | \$25 |
| | PRO Survey #1 | \$25 |
| Month 12 | PRO Survey #2 | \$30 |

## **Incentive Mapping for Oral PrEP Arm**

| Time Frame | Activity | Incentive |
|------------|-----------------------------|-----------|
| Month 0 | Baseline Demographic Survey | \$20 |
| Month 1 | Persistence assessment | \$5 |
| | PRO Survey #1 | \$10 |
| Month 2 | Health Literacy Survey | \$5 |
| | Persistence assessment | \$5 |
| Month 3 | PRO Survey #2 | \$10 |
| | Persistence assessment | \$10 |
| Month 4 | Health Literacy Survey | \$5 |
| | Persistence assessment | \$10 |
| Month 5 | Persistence assessment | \$10 |
| | PRO Survey #1 | \$10 |
| Month 6 | Health Literacy Survey | \$5 |
| | Persistence assessment | \$10 |
| Month 7 | Persistence assessment | \$10 |
| Month 8 | Health Literacy Survey | \$5 |
| | Persistence assessment | \$10 |
| Month 9 | PRO Survey #2 | \$15 |
| | Persistence assessment | \$15 |
| Month 10 | Health Literacy Survey | \$5 |
| | Persistence assessment | \$15 |
| Month 11 | Persistence assessment | \$15 |
| | PRO Survey #1 | \$20 |
| Month 12 | Persistence assessment | \$15 |
| | PRO Survey #2 | \$25 |

### Appendix F: Overview of TheraPay App Screens for Aurora PrEP Study

# WVHR CAB LA PrEP DEMO 2023 Screenshots



Opening Screen (this is the first screen members see after going through the sign-up process)



Multiple Plan Carousel screen shows the different Plans for which a Highmark Healthy

Rewards member is enrolled, the number of activities in the Plan, and
the total rewards available in the Plan.



Health Right. | PR INTE

Overview screen shows all tasks each person is eligible within each plan, examples of the tasks in each plan are in the screenshots below. Tasks that have expired are marked by a red "x", tasks that are open have an open check box, tasks that are still locked have a padlock image.



Up Next shows you only the open tasks, or in other words, all the activities that are available for you to complete now. Tasks will open on certain dates, or when previous tasks are completed that unlock the next task.



When members tap either the circles (in the Overview page) or the tiles (in the Up Next page), each one comes with more details. The screens below are for those pages.











In the My Money section, the member can see what their balance is on their card, any transactions from their card, and any special offers available to them.



The My Progress Page shows how much progress a member has made against their activities and how much is still available.



## Generic Push Notifications identify accomplishments, validations, and funds received.



#### Appendix G: Study Schema

Patients >18 y/o who are newly started on PrEP therapy at WVHR and have access to a smart phone with data (N=105)

- V. Participants will have been prescribed CAB-LA, daily FTC/TDF, or daily FTC/TAF in accordance with the WVHR standard of care by a licensed HCP prior to enrolling in the study
- VI. Not receiving HIV PrEP care outside of WVHR
- VII. No positive HIV diagnosis
- VIII. No contraindications to oral or injectable PrEP therapy

# CAB-LA PrEP Arm n = 70

- PrEP injections at months0, 1, 3, 5, 7, 9 and 11
- Education modules at months 2, 4, 6, 8, and 10

## Oral PrEP Arm n = 35

- PrEP prescription fills at months0, 3, 6, 9, and 12
- Education modules at months 2, 4, 6, 8, and 10

**Primary outcome measure:** mean patient-reported adherence and persistence at months 3 and end of study, validated by medication ratio between the CAB-LA and Oral Prep cohorts

**Secondary outcome measure 1**: retention in care in patients receiving CAB-LA vs oral PrEP defined as the proportion of patients presenting for their follow-up appointments within 30 days of their scheduled visit at months 3, 9 and 12 for the Oral PrEP cohort and at months 3, 9, and 11 for the CAB-LA cohort

**Secondary outcome measure 2:** patient-reported outcomes including PrEP medication satisfaction, PrEP acceptance, and PrEP-related stigma, and barriers to adherence and reasons for PrEP discontinuation assessed through brief behavioral surveys

**Secondary outcome measure 3**: implementation outcomes including patient acceptability (AIM), appropriateness (IAM), and helpfulness of the education modules within the digital health program assessed using a Likert scale and health literacy evaluation

**Secondary outcome measure 4:** clinician acceptability, appropriateness, and feasibility of implementing long-acting cabotegravir injections (AIM, IAM, FIM), and barriers to and facilitators for implementation of CAB-LA

Appendix H: Study Timelines

| CAB-LA PrEP Arm (N=70) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month 0 | Month 0 | Month 1 | Month 2 | Month 3 | Month 4 | Month 5 | Month 6 | Month 7 | Month 8 | Month 9 | Month 10 | Month 11 | Month 12 |
| Baseline labs<br>and<br>1st PrEP<br>injection<br>Baseline<br>demographic<br>survey | Baseline<br>evaluation<br>and<br>introduction<br>to support<br>group | 2nd PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection—<br>Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>3rd PrEP<br>injection<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>4th PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection—<br>Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>5th PrEP<br>injection<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>6th PFEP<br>injection<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation | Follow-up<br>labs and<br>7th PrEP<br>injection<br>Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | PRO data<br>collection –<br>Set #2 |
| Oral PrEP Arm (N=35) | | | | | | | | | | | | | |
| Month 0 | Month 0 | Month 1 | Month 2 | Month 3 | Month 4 | Month 5 | Month 6 | Month 7 | Month 8 | Month 9 | Month 10 | Month 11 | Month 12 |
| Baseline labs<br>and<br>PrEP<br>prescription<br>filled<br>Baseline<br>demographic<br>survey | Baseline<br>evaluation<br>and<br>introduction<br>to support<br>group | Persistence<br>Assessment PRO data<br>collection – Set #1 | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Follow-up<br>labs and<br>PrEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Follow-up<br>labs and<br>PFEP<br>prescription<br>refill<br>Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Follow-up<br>labs and<br>PrEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment | Education<br>modules and<br>health<br>literacy<br>evaluation<br>Persistence<br>Assessment | Persistence<br>Assessment<br>PRO data<br>collection –<br>Set #1 | Follow-up<br>labs and<br>PrEP<br>prescription<br>refill<br>PRO data<br>collection –<br>Set #2<br>Persistence<br>Assessment |
| Reciprocity App – Education Modules Month 2: PrEP Medicines Month 4:Protecting Yourself from HIV, STIs, and other infections Month 6: Building a Support System for HIV Prevention Month 8: Being an Active Participant in Your Own Care Month 10: Overcoming Stigma and Becoming a Health Advocate | | | | | | PrEP Medication Satisfaction PrEP-Related Stigma PrEP Acceptance IAM | | | | | | | |

| Clinic St | taff | | | | | | | | | | | | | | End of Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month 0 | Month 0 | Month 1 | Month 2 | Month 3 | Month 4 | Month 5 | Month 6 | Month 7 | Month 8 | Month 9 | Month 10 | Month 11 | Month 12 | | Liid oi Study |
| | | | | | | | | | | | | | | | AIM, IAM, FIM, |
| Baseline<br>Provider | AIM, IAM,<br>FIM | | | | | | AIM, IAM,<br>FIM, Follow-<br>Up Provider | | | | | | AIM, IAM,<br>FIM, Follow-<br>Up, Provider | 7 | Follow-up |
| Survey | | | | | | | Survey | | | | | | Survey | | Provider Survey |

### Appendix I: Forms for Safety Reporting

WV HealthRight will use GSK/ViiV reporting forms (for SAE, medical device incident and pregnancies. Completed forms will be sent to the GSK PV Operations group.

### **SAFETY DATA EXCHANGE**

### Adverse Event and Serious Adverse Event Definitions

For the purposes of this Agreement, an Adverse Event (AE) shall mean any untoward medical occurrence whether thought to have been caused by the ViiV IMP or the Study or not, and a Serious Adverse Event (SAE) shall mean any adverse event which is fatal, life threatening, disabling or incapacitating, requires in-patient treatment or prolongs existing hospitalization, is a congenital anomaly in the off-spring of the patient or which may require intervention to prevent the previously stated outcomes.

### Medical Device Incident Definition

For the purposes of this Agreement a medical device incident is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Device incidents include malfunctions, use errors, and/or deficiencies of the information supplied by the manufacturer. Device deficiencies/incidents may result in an SAE (including death or serious deterioration in health of a subject, or other non-participant person) or a non-serious AE, or lead to an SAE or AE if appropriate action had not been taken or, intervention had not occurred. The requirement to report medical device incidents applies to any incident occurring in association with a medical device provided in a ViiV commercial pack for the ViiV IMP(s) or any other known ViiV medicinal product.

### Reporting Clinical Safety Information to GSK on behalf of ViiV

The Sponsor shall require the Participating Institution to report all Serious Adverse Events, Pregnancy Exposures and Medical Device Incidents disclosed by Study Subjects, or identified from review of Medical Records/Questionnaires during the course of the Study, for which the Participating Institution considers there to be a reasonable possibility of causal relationship with the ViiV IMP or any other known ViiV Product within 24 hours of first becoming aware of the event, regardless of Sponsor/designee expectedness assessments. Sponsor shall require of Participating Institutions that if the Participating Institution is unable to confirm whether ViiV is the manufacturer of the relevant product, Participating Institution shall nonetheless report the event to ViiV.

### Routing of Clinical Safety Data to GSK

Notwithstanding Section 23 ['NOTICES'] of the Agreement, such reports and information as outlined above, including Investigator causality assessments against all concerned ViiV Products(s) and English translations of all information where reporting is from a non-English speaking country, shall be sent to the: GSK PV Operations Group at email: OAX37649@gsk.com OR if Sponsor is unable to email the report, Sponsor may send the report via facsimile

number+44-208 1814780. Should SPONSOR experience difficulty submitting a report, contact the ViiV individual listed in Section 23 "Notices".

### Requesting Follow up information:

The Sponsor shall require the Participating Institution to provide GSK's safety department with details of whom GSK or ViiV shall address requests for follow up information from this Study, and further agrees to update such contact details as necessary. At the time of this Agreement, all such requests should be addressed to: David Hardy wdavidhardymd@gmail.com Sponsor shall require the Participating Institution shall submit to GSK (as specified above) such further detailed information relating there to as GSK shall request within 24 hours of it becoming available.